CLINICAL TRIAL: NCT00121641
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Trial to Evaluate the Efficacy and Safety of Saxagliptin (BMS-477118) as Monotherapy in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control With Diet and Exercise
Brief Title: Saxagliptin Treatment in Subjects With Type 2 Diabetes Who Are Not Controlled With Diet and Exercise
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-011
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Results first posted 2011-05-11 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (5):
- Saxagliptin 2.5 mg (A) (Experimental): Metformin 500-2000 mg (as needed for rescue)
  Interventions: Drug: Saxagliptin; Drug: Placebo matching Metformin; Drug: Metformin
- Saxagliptin 5 mg (B) (Experimental): Metformin 500-2000 mg (as needed for rescue)
  Interventions: Drug: Saxagliptin; Drug: Placebo matching Metformin; Drug: Metformin
- Saxagliptin 10 mg (C) (Experimental): Metformin 500-2000 mg (as needed for rescue)
  Interventions: Drug: Saxagliptin; Drug: Placebo matching Metformin; Drug: Metformin
- Placebo (D) (Placebo Comparator): Metformin 500-2000 mg (as needed for rescue)
  Interventions: Drug: Placebo matching Saxagliptin; Drug: Metformin
- Open-Label Treatment Cohort (Direct Enrollees) (E) (Experimental): Saxagliptin 10 mg
  Metformin 500-2000 mg (as needed for rescue)
  Interventions: Drug: Saxagliptin; Drug: Metformin

INTERVENTIONS:
Drug: Saxagliptin — Tablets, Oral, 2.5 mg, Once daily (24 weeks short term [ST], 42 months long term [LT])
  Other Names: BMS-477118
  Arms: Saxagliptin 2.5 mg (A)
Drug: Saxagliptin — Tablets, Oral, 5 mg, Once daily (24 weeks ST, 42 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin 5 mg (B)
Drug: Saxagliptin — Tablets, Oral, 10 mg, Once daily (24 weeks ST, 42 months LT)
  Other Names: BMS-477118
  Arms: Saxagliptin 10 mg (C)
Drug: Placebo matching Saxagliptin — Tablets, Oral, 0mg, Once daily (24 weeks ST, 42 months LT)
  Arms: Placebo (D)
Drug: Metformin — Tablets, Oral, 500 mg, daily (42 months LT)
  Arms: Placebo (D)
Drug: Placebo matching Metformin — Tablets, Oral, 0 mg, daily (42 months LT)
  Arms: Saxagliptin 10 mg (C); Saxagliptin 2.5 mg (A); Saxagliptin 5 mg (B)
Drug: Saxagliptin — Tablets, Oral, 10 mg, Once daily (24 weeks ST, 42 months LT) Open Label
  Other Names: BMS-477118
  Arms: Open-Label Treatment Cohort (Direct Enrollees) (E)
Drug: Metformin — Tablets, Oral, 500-2000 mg (as needed for rescue)

SUMMARY:
The purpose of this clinical research study is to learn whether saxagliptin (BMS-477118) is more effective than placebo as a treatment for type 2 diabetic subjects who are not sufficiently controlled with diet and exercise

DETAILED DESCRIPTION:
All subjects will participate in a lead-in period, and qualifying subjects will continue into a short-term randomized treatment period. Subjects who complete the short-term period will be eligible to enter the long term extension period. Also, subjects in the short-term period who have an elevated blood sugar that requires additional medication for blood sugar control will be eligible to enter the long-term treatment extension period where they will receive metformin added onto their blinded study medication. Subjects with screening hemoglobin A1c (A1C) > 10.0% and ≤ 12.0%, who otherwise meet all inclusion/exclusion criteria, were eligible to enroll directly into Open-Label Treatment Cohort (Direct Enrollees) and receive open-label saxagliptin 10 mg. Those who completed the short-term period were eligible to enter into the long-term treatment extension period.Saxagliptin dose titration was not permitted.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Drug naive
* Hemoglobin (Hb) A1c >= 7.0% and <= 10.0% (>10% and <= 12% for open label arm)
* Fasting C-peptide >= 1 ng/mL
* Body mass index <= 40 kg/m2

Exclusion Criteria:

* Symptomatic poorly controlled diabetes
* Recent cardiac or cerebrovascular event
* Serum creatinine >= 1.5 mg/dL for males and >= 1.4 mg/dL for Women of Child Bearing Potential

Ages: 18 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1035 (Actual)
Dates: Start 2005-07; Primary Completion 2006-08 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (134):
- United States (83):
  - Local Institution, Anniston, Alabama
  - Local Institution, Birmingham, Alabama
  - Local Institution, Calera, Alabama
  - Local Institution, Jonesboro, Arizona
  - Local Institution, Mesa, Arizona
  - Local Institution, Pheonix, Arizona
  - Local Institution, Little Rock, Arkansas
  - Local Institution, Anaheim, California
  - Local Institution, Fountain Valley, California
  - Local Institution, Fresno, California
  - Local Institution, Long Beach, California
  - Local Institution, Los Angeles, California
  - Local Institution, Northridge, California
  - Local Institution, Rolling Hills Estates, California
  - Local Institution, Sacramento, California
  - Local Institution, Santa Ana, California
  - Local Institution, Spring Valley, California
  - Local Institution, Tustin, California
  - Local Institution, Castle Rock, Colorado
  - Local Institution, Denver, Colorado
  - Local Institution, Loveland, Colorado
  - Local Institution, Altamonte Springs, Florida
  - Local Institution, Chipley, Florida
  - Local Institution, Cocoa Beach, Florida
  - Local Institution, Coral Gables, Florida
  - Local Institution, Fort Lauderdale, Florida
  - Local Institution, Jupiter, Florida
  - Local Institution, Kissimmee, Florida
  - Local Institution, Marianna, Florida
  - Local Institution, New Port Richey, Florida
  - Local Institution, Ocala, Florida
  - Local Institution, West Palm Beach, Florida
  - Local Institution, Vernon Hills, Illinois
  - Local Institution, Dubuque, Iowa
  - Local Institution, Iowa City, Iowa
  - Local Institution, Waterloo, Iowa
  - Local Institution, Wichita, Kansas
  - Local Institution, Lexington, Kentucky
  - Local Institution, Munfordville, Kentucky
  - Local Institution, New Orleans, Louisiana
  - Local Institution, West Monroe, Louisiana
  - Local Institution, Baltimore, Maryland
  - Local Institution, Chester, Maryland
  - Local Institution, Prince Frederick, Maryland
  - Local Institution, Ayer, Massachusetts
  - Local Institution, Boston, Massachusetts
  - Local Institution, Rolling Fork, Mississippi
  - Local Institution, Kansas City, Missouri
  - Local Institution, Springfield, Missouri
  - Local Institution, St Louis, Missouri
  - Local Institution, Kalispell, Montana
  - Local Institution, Omaha, Nebraska
  - Local Institution, Las Vegas, Nevada
  - Local Institution, Middletown, New Jersey
  - Local Institution, Toms River, New Jersey
  - Local Institution, Cooperstown, New York
  - Local Institution, Greensboro, North Carolina
  - Local Institution, Huntersville, North Carolina
  - Local Institution, Sparta, North Carolina
  - Local Institution, Statesville, North Carolina
  - Local Institution, Winston-Salem, North Carolina
  - Local Institution, Athens, Ohio
  - Local Institution, Franklin, Ohio
  - Local Institution, Oklahoma City, Oklahoma
  - Local Institution, Tulsa, Oklahoma
  - Local Institution, Portland, Oregon
  - Local Institution, Fleetwood, Pennsylvania
  - Local Institution, Philadelphia, Pennsylvania
  - Local Institution, Pittsburgh, Pennsylvania
  - Local Institution, Charleston, South Carolina
  - Local Institution, Bristol, Tennessee
  - Local Institution, Morristown, Tennessee
  - Local Institution, Bryan, Texas
  - Local Institution, Dallas, Texas
  - Local Institution, Fort Worth, Texas
  - Local Institution, Houston, Texas
  - Local Institution, San Antonio, Texas
  - Local Institution, Temple, Texas
  - Local Institution, Texarkana, Texas
  - Local Institution, The Colony, Texas
  - Local Institution, Salt Lake City, Utah
  - Local Institution, Virginia Beach, Virginia
  - Local Institution, Olympia, Washington
- Australia (8):
  - Local Institution, Sydney, New South Wales
  - Local Institution, Woollongong, New South Wales
  - Local Institution, Brisbane, Queensland
  - Local Institution, Kippa-Ring, Queensland
  - Local Institution, Meadowbrook, Queensland
  - Local Institution, Adelaide, South Australia
  - Local Institution, Woodville South, South Australia
  - Local Institution, Perth, Western Australia
- Canada (29):
  - Local Institution, Calgary, Alberta
  - Local Institution, Edmonton, Alberta
  - Local Institution, Kelowna, British Columbia
  - Local Institution, Quesnel, British Columbia
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Portage la Prairie, Manitoba
  - Local Institution, Winnipeg, Manitoba
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, Moncton, New Brunswick
  - Local Institution, Manuels, Newfoundland and Labrador
  - Local Institution, Mount Pearl, Newfoundland and Labrador
  - Local Institution, St. John's, Newfoundland and Labrador
  - Local Institution, Newmarket, Ontario
  - Local Institution, Oakville, Ontario
  - Local Institution, Peterborough, Ontario
  - Local Institution, Sarnia, Ontario
  - Local Institution, Strathroy, Ontario
  - Local Institution, Thornhill, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Drummondville, Quebec
  - Local Institution, Fleurimont, Quebec
  - Local Institution, Gatineau, Quebec
  - Local Institution, Granby, Quebec
  - Local Institution, Longueuil, Quebec
  - Local Institution, Montreal, Quebec
  - Local Institution, Saint-Léonard, Quebec
  - Local Institution, Ste-Foy, Quebec
  - Local Institution, Saskatoon, Saskatchewan
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Durango, Durango
  - Local Institution, Guadalajara, Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Hermosillo, Sonora
- Puerto Rico (5):
  - Local Institution, Carolina
  - Local Institution, Guaynabo
  - Local Institution, Ponce
  - Local Institution, Rio Piedras
  - Local Institution, San Juan
- Taiwan (3):
  - Local Institution, Hualien City
  - Local Institution, Taichung
  - Local Institution, Taipei

REFERENCES:
- [Background] Rosenstock J, Aguilar-Salinas C, Klein E, Nepal S, List J, Chen R; CV181-011 Study Investigators. Effect of saxagliptin monotherapy in treatment-naive patients with type 2 diabetes. Curr Med Res Opin. 2009 Oct;25(10):2401-11. doi: 10.1185/03007990903178735. PMID 19650754
- [Derived] Esu E, Berens-Riha N, Pritsch M, Nwachuku N, Loescher T, Meremikwu M. Intermittent screening and treatment with artemether-lumefantrine versus intermittent preventive treatment with sulfadoxine-pyrimethamine for malaria in pregnancy: a facility-based, open-label, non-inferiority trial in Nigeria. Malar J. 2018 Jul 6;17(1):251. doi: 10.1186/s12936-018-2394-2. PMID 29976228
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391
- [Derived] Bonora E, Bryzinski B, Hirshberg B, Cook W. A post hoc analysis of saxagliptin efficacy and safety in patients with type 2 diabetes stratified by UKPDS 10-year cardiovascular risk score. Nutr Metab Cardiovasc Dis. 2016 May;26(5):374-9. doi: 10.1016/j.numecd.2015.11.004. Epub 2015 Dec 1. PMID 27033025
- [Derived] Rosenstock J, Gross JL, Aguilar-Salinas C, Hissa M, Berglind N, Ravichandran S, Fleming D. Long-term 4-year safety of saxagliptin in drug-naive and metformin-treated patients with Type 2 diabetes. Diabet Med. 2013 Dec;30(12):1472-6. doi: 10.1111/dme.12267. Epub 2013 Jul 19. PMID 23802840

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1035 subjects were enrolled; 422 entered the 2-week dietary/exercise placebo lead-in. 21 did not enter double-blind treatment period (19 discontinued, 2 randomized but did not receive study drug). 68 with screening hemoglobin A1c (A1C) >10.0% and ≤12.0% entered directly in the open-label cohort; 66 received at least 1 dose of saxagliptin 10mg.
Groups:
- Saxagliptin 2.5 mg: Tablets, Oral, 2.5 mg, Once daily (24 weeks short term [ST], 42 months long term [LT]); Metformin 500-2000 mg (as needed for rescue).
- Saxagliptin 5 mg: Tablets, Oral, 5 mg, Once daily (24 weeks ST, 42 months LT); Metformin 500-2000 mg (as needed for rescue).
- Saxagliptin 10 mg; Open-Label Treatment Cohort (Direct Enrollees): Tablets, Oral, 10 mg, Once daily (24 weeks ST, 42 months LT); Metformin 500-2000 mg (as needed for rescue).
- Placebo: Tablets, Oral, 0mg, Once daily (24 weeks ST, 42 months LT); Metformin 500-2000 mg (as needed for rescue)
Period: 24-week Short-term Treatment Period
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo | Open-Label Treatment Cohort (Direct Enrollees)
Started | 102 | 106 | 98 | 95 | 66
Completed | 73 | 68 | 69 | 55 | 25
Not Completed | 29 | 38 | 29 | 40 | 41
Not completed — Lack of Efficacy | 15 | 21 | 14 | 25 | 30
Not completed — Subject Withdrew Consent | 9 | 11 | 5 | 10 | 3
Not completed — Adverse Event | 3 | 3 | 4 | 0 | 2
Not completed — Lost to Follow-up | 0 | 2 | 3 | 4 | 4
Not completed — Poor / Non-compliance | 0 | 0 | 3 | 1 | 1
Not completed — Subject No Longer Meets Study Criteria | 1 | 1 | 0 | 0 | 1
Not completed — Other Reason | 1 | 0 | 0 | 0 | 0
Period: 48-month Short Term + Long Term Period
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo | Open-Label Treatment Cohort (Direct Enrollees)
Started | 102 | 106 | 98 | 95 | 66
Completed | 23 | 24 | 28 | 24 | 8
Not Completed | 79 | 82 | 70 | 71 | 58
Not completed — Lack of Efficacy | 26 | 27 | 21 | 26 | 25
Not completed — Subject Withdrew Consent | 25 | 28 | 17 | 24 | 10
Not completed — Adverse Event | 9 | 10 | 10 | 5 | 5
Not completed — Lost to Follow-up | 9 | 7 | 12 | 11 | 12
Not completed — Poor / Non-compliance | 4 | 1 | 4 | 2 | 2
Not completed — Subject No Longer Meets Study Criteria | 1 | 3 | 2 | 1 | 2
Not completed — Pregnancy | 0 | 1 | 0 | 1 | 0
Not completed — Administrative Reason by Sponsor | 0 | 2 | 1 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 1 | 0
Not completed — Missing | 0 | 0 | 1 | 0 | 0
Not completed — Other Reason | 5 | 3 | 2 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Saxagliptin 2.5 mg: Tablets, Oral, 2.5 mg, Once daily (24 weeks ST, 42 months LT); Metformin 500-2000 mg (as needed for rescue).
- Total: Total of all reporting groups
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo | Total
Number analyzed (Participants) | 102 | 106 | 98 | 95 | 401
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.27 (10.06) | 53.91 (11.57) | 52.73 (11.27) | 53.91 (12.32) | 53.46 (11.29)
Age, Customized [Number; unit: participants]
  <65 years | 91 | 86 | 84 | 77 | 338
  >= 65 years | 11 | 20 | 14 | 18 | 63
  >=75 years | 2 | 1 | 1 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 52 | 53 | 48 | 197
  Male | 58 | 54 | 45 | 47 | 204
Race/Ethnicity, Customized [Number; unit: participants]
  White | 89 | 93 | 80 | 79 | 341
  Black/African American | 5 | 5 | 6 | 6 | 22
  Asian | 5 | 4 | 6 | 3 | 18
  Other | 3 | 4 | 6 | 7 | 20
  Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Partcipants]
  Hispanic / Latino | 16 | 14 | 14 | 15 | 59
  Not Hispanic / Latino | 45 | 49 | 42 | 38 | 174
  Not Reported | 41 | 43 | 42 | 42 | 168
Age Categorization, Female Only [Number; unit: Participants]
  =< 50 years | 17 | 24 | 22 | 19 | 82
  > 50 years | 27 | 28 | 31 | 29 | 115
Weight [Mean (Standard Deviation); unit: kg] | 92.10 (18.39) | 91.09 (18.53) | 89.30 (17.67) | 86.56 (16.90) | 89.84 (17.96)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.90 (4.82) | 32.30 (4.53) | 31.71 (4.71) | 30.93 (4.26) | 31.73 (4.60)
Body Mass Index Categorization [Number; unit: Participants]
  < 30 | 36 | 40 | 35 | 42 | 153
  >= 30 | 66 | 66 | 63 | 53 | 248

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c (A1C) Changes From Baseline at Week 24
Description: To compare the change from baseline in HbA1c achieved with each dose of saxagliptin versus placebo in treatment naive subjects with type 2 diabetes who have inadequate glycemic control defined as A1C ≥7.0% and ≤10.0%.
Time Frame: Baseline, Week 24
Population: Randomized participants with both a baseline and post-baseline value (up to Week 24).
Measure: Mean (Standard Error); unit: Percentage of glycosylated hemoglobins
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
Percentage of glycosylated hemoglobins
  Baseline Mean | 7.91 (0.09) | 7.98 (0.11) | 7.85 (0.09) | 7.88 (0.10)
  Adjusted Mean Change from Baseline | -0.43 (0.10) | -0.46 (0.10) | -0.54 (0.10) | 0.19 (0.10)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg vs Placebo; Test type: Superiority or Other; p < .0001, ANCOVA — Between-group comparisons significant at alpha = 0.019, significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -0.62, 95% CI 2-sided [-0.90 to -0.33], Standard Error of Mean 0.14 — ANCOVA model:post - pre = pre treatment
Statistical Analysis 2: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p < .0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -0.64, 95% CI 2-sided [-0.93 to -0.36], Standard Error of Mean 0.14 — ANCOVA model:post - pre = pre treatment
Statistical Analysis 3: Comparison: Saxagliptin 10 mg vs Placebo; Test type: Superiority or Other; p < .0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -0.73, 95% CI 2-sided [-1.02 to -0.44], Standard Error of Mean 0.15 — ANCOVA model:post - pre = pre treatment

2. Secondary Outcome: Baseline and Change From Baseline at Week 24 in Fasting Plasma Glucose (FPG)
Time Frame: Baseline, Week 24
Population: Randomized participants with measure at given time points, Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 101 | 105 | 97 | 92
mg/dL
  Baseline | 177.72 (4.12) | 171.31 (4.09) | 176.51 (4.43) | 171.85 (4.80)
  Adjusted Change from Baseline | -14.53 (3.82) | -8.67 (3.74) | -16.75 (3.89) | 6.06 (4.00)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -20.60, 95% CI 2-sided [-31.47 to -9.72], Standard Error of Mean 5.53 — ANCOVA model:post - pre = pre treatment
Statistical Analysis 2: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.0074, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -14.73, 95% CI 2-sided [-25.50 to -3.97], Standard Error of Mean 5.48 — ANCOVA model:post - pre = pre treatment
Statistical Analysis 3: Comparison: Saxagliptin 10 mg vs Placebo; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -22.81, 95% CI 2-sided [-33.79 to -11.84], Standard Error of Mean 5.58 — ANCOVA model:post - pre = pre treatment

3. Secondary Outcome: Percentage of Participants Achieving Therapeutic Glycemic Response (A1C < 7.0%) at Week 24
Time Frame: Week 24
Population: Randomized Participants with measurement at time point, Last Observation Carried Forward (LOCF)
Measure: Number; unit: percentage of participants
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 100 | 103 | 95 | 92
percentage of participants | 35.0 | 37.9 | 41.1 | 23.9
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.1141, Fisher Exact — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; The exact 95% CIs is based on the standardized statistic and inverting the one 2-sided test; Difference in Proportions = 11.1, 95% CI 2-sided [-3.1 to 24.9]
Statistical Analysis 2: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.0443, Fisher Exact — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; The exact 95% CIs is based on the standardized statistic and inverting the one 2-sided test; Difference in Proportions = 14.0, 95% CI 2-sided [-0.1 to 27.6]
Statistical Analysis 3: Comparison: Saxagliptin 10 mg vs Placebo; Test type: Superiority or Other; p = 0.0133, Fisher Exact — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; The exact 95% CIs is based on the standardized statistic and inverting the one 2-sided test; Difference in Proportions = 17.1, 95% CI 2-sided [2.8 to 31.0]

4. Secondary Outcome: Baseline and Change From Baseline at Week 24 in Postprandial Glucose (PPG) Area Under the Curve (AUC)
Time Frame: Baseline, Week 24
Population: Randomized participants with measure at given time points, Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 74 | 79 | 73 | 66
mg*min/dL
  Baseline | 45030 (1368.1) | 45691 (1209.8) | 44614 (1394.0) | 46030 (1397.8)
  Adjusted Change from Baseline | -6868 (1167.7) | -6896 (1130.2) | -8084 (1176.2) | -646.6 (1236.9)
Statistical Analysis 1: Comparison: Saxagliptin 2.5 mg vs Placebo; Test type: Superiority or Other; p = 0.0003, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -6221, 95% CI 2-sided [-9570 to -2872], Standard Error of Mean 1701.3 — ANCOVA model:post - pre = pre treatment
Statistical Analysis 2: Comparison: Saxagliptin 5 mg vs Placebo; Test type: Superiority or Other; p = 0.0002, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -6249, 95% CI 2-sided [-9546 to -2952], Standard Error of Mean 1675.1 — ANCOVA model:post - pre = pre treatment
Statistical Analysis 3: Comparison: Saxagliptin 10 mg vs Placebo; Test type: Superiority or Other; p < .0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -7437, 95% CI 2-sided [-10798 to -4076], Standard Error of Mean 1707.6 — ANCOVA model:post - pre = pre treatment

5. Secondary Outcome: Baseline and Change From Baseline at Week 24 in Fasting Plasma Glucose (FPG) - Open Label Cohort
Time Frame: Baseline, Week 24
Population: Open Label Subjects with Measurement at Timepoint; Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- Open-Label Cohort (Direct Enrollees): Tablets, Oral, 10 mg, Once daily (24 weeks ST, 42 months LT); Metformin 500-2000 mg (as needed for rescue).
Arm/Group | Open-Label Cohort (Direct Enrollees)
Number analyzed (Participants) | 64
mg/dL
  Baseline | 241.08 (6.19)
  Change from Baseline | -33.42 (5.37)

6. Secondary Outcome: Percentage of Participants Achieving Therapeutic Glycemic Response (A1C < 7.0%) at Week 24 - Open Label Cohort
Time Frame: Week 24
Population: Open Label Participants with measurement at time point, Last Observation Carried Forward (LOCF)
Measure: Number; unit: percentage of participants
Groups:
- Open Label Cohort (Direct Enrollees): Tablets, Oral, 10 mg, Once daily (24 weeks ST, 42 months LT); Metformin 500-2000 mg (as needed for rescue).
Arm/Group | Open Label Cohort (Direct Enrollees)
Number analyzed (Participants) | 64
percentage of participants | 14.1

7. Primary Outcome: A1C Changes From Baseline at Week 24 - Open Label Cohort
Description: as for outcome 1
Time Frame: Baseline, Week 24
Population: Open-label participants with both a baseline and a post-baseline (up to Week 24)
Measure: Mean (Standard Error); unit: Percentage of glycosylated hemoglobins
Arm/Group | Open Label Cohort (Direct Enrollees)
Number analyzed (Participants) | 64
Percentage of glycosylated hemoglobins
  Baseline Mean | 10.70 (0.10)
  Mean Change from Baseline | -1.87 (0.18)

8. Secondary Outcome: Baseline and Change From Baseline at Week 24 in Postprandial Glucose (PPG) Area Under the Curve (AUC) - Open Label Cohort
Time Frame: Baseline, Week 24
Population: Open Label participants with measure at given time points, Last Observation Carried Forward (LOCF).
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Open Label Cohort (Direct Enrollees)
Number analyzed (Participants) | 64
mg*min/dL
  Baseline | 60687 (2312.4)
  Change from Baseline | -11078 (2132.8)

9. Other Pre Specified Outcome: Baseline Demographic Characteristic (Age, Continuous) - Summary for ST + LT Treatment Period - Open-Label Cohort
Description: This cohort represents a different population (screening A1C > 10.0% and ≤ 12.0%) than the double-blind cohort, and was presented separately in the study report.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
years | 49.09 (8.63)

10. Other Pre Specified Outcome: Baseline Demographic Characteristics - Summary for ST + LT Treatment Period - Open-Label Cohort
Description: as for outcome 9
Time Frame: Baseline
Measure: Number; unit: participants
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
participants
  Age <65 years | 64
  Age >=65 years | 2
  Age >=75 years | 0
  Gender, Male | 32
  Gender, Female | 34
  Age =<50 years, females only | 19
  Age >50 years, females only | 15
  Race, White | 61
  Race, Black/African American | 3
  Race, Asian | 1
  Race, Other | 1
  Ethnicity, Hispanic/Latino | 13
  Ethnicity, Not Hispanic/Latino | 37
  Ethnicity, Not Reported | 16
  Body Mass Index <30% | 22
  Body Mass Index >=30% | 44

11. Other Pre Specified Outcome: Baseline Demographic Characteristic (Weight) - Summary for ST + LT Treatment Period - Open-Label Cohort
Description: as for outcome 9
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
kg | 91.41 (20.65)

12. Other Pre Specified Outcome: Baseline Demographic Characteristic (Body Mass Index) - Summary for ST + LT Treatment Period - Open-Label Cohort
Description: as for outcome 9
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
kg/m^2 | 31.73 (4.73)

13. Other Pre Specified Outcome: Overall Summary of Adverse Events During ST+LT Treatment Period
Description: AE=any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with this treatment. SAE=any untoward medical occurrence that at any dose: results in death, is life-threatening, requires inpatient hospitalization or causes prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, results in development of drug dependency or drug abuse, is an important medical event. Related events=relationship of certain, probable, possible, or missing.
Time Frame: AEs: up to last treatment day + 1 day or last visit; SAEs: up to last treatment day + 30 days or last visit + 30 days. Mean duration of exposure was 109 weeks in 10 mg arm, 94.7 weeks in 2.5 mg arm, 103 weeks in 5 mg arm, and 98.4 weeks in placebo arm.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
participants
  At Least 1 AE | 89 | 94 | 87 | 77
  At Least 1 Related AE | 25 | 23 | 25 | 25
  Deaths | 0 | 0 | 0 | 1
  At Least 1 SAE | 11 | 18 | 9 | 11
  At Least 1 Related SAE | 0 | 1 | 0 | 0
  Discontinuations Due to SAEs | 6 | 2 | 3 | 1
  Discontinuations Due to AEs | 9 | 10 | 10 | 5

14. Other Pre Specified Outcome: Marked Laboratory Abnormalities - During ST + LT Treatment Period
Description: A laboratory value was considered a marked abnormality if it is outside the pre-defined criteria for marked abnormality and the on-treatment value was more extreme (farther from the limit) than the baseline value. Pre-Rx=pretreatment; ULN=upper limit of normal; ALP=alkaline phosphatase; AST=aspartate aminotransferase; ALT=alanine aminotransferase; unspec=unspecified; sodium serum low: <0.9 x Pre-Rx & <=130mEq/L / high: >1.1 x Pre-Rx & >=150mEq/L; potassium, serum low: <=0.8 x Pre-Rx & >=6.0mEq/L / high: 1.2 x Pre-Rx & >=6.0mEq/L; LLN=lower limit of normal.
Time Frame: Lab assessments taken during and up to 14 days after the last dose of study drug during the ST + LT Treatment Period. Mean duration of exposure was 109 weeks in 10 mg arm, 94.7 weeks in 2.5 mg arm, 103 weeks in 5 mg arm, and 98.4 weeks in placebo arm.
Population: Number of Participants Analyzed=Treated participants; n=number of treated subjects with baseline value and at least one value during the ST + LT treatment period
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
participants
  Hemoglobin < 8 g/dL (n=101, 105, 97, 93) | 0 | 0 | 0 | 0
  Hematocrit < 0.75 x pre-Rx (n=101, 105, 97, 93) | 0 | 0 | 1 | 0
  Platelets < 50 x 10^9 c/L (n=100, 104, 94, 93) | 0 | 0 | 0 | 0
  Platelets > 1.5 x ULN (n=100,104, 94, 93) | 1 | 0 | 0 | 1
  Leukocytes < 2 x 1000 c/µL (n=101, 105, 97, 93) | 0 | 0 | 0 | 0
  Neutrophils+Bands <1x1000 c/µL(n=101, 105, 97, 93) | 0 | 0 | 1 | 0
  Eosinophils >0.9x1000 c/µL (n=101, 105, 97, 93) | 1 | 5 | 3 | 4
  Lymphocytes <=0.75x1000 c/µL (n=101, 105, 97, 93) | 4 | 2 | 2 | 1
  ALP >3 x pre-Rx and >ULN (n=101,105, 97, 94) | 0 | 0 | 0 | 0
  ALP >1.5 x ULN (n=101, 105, 97, 94) | 2 | 1 | 1 | 1
  AST >3 x ULN (n=101, 105, 97, 94) | 3 | 2 | 1 | 0
  AST >5 x ULN (n=101, 105, 97, 94) | 2 | 1 | 0 | 0
  AST >10 x ULN (n=101, 105, 97, 94) | 1 | 0 | 0 | 0
  AST >20 x ULN (n=101, 105, 97, 94) | 0 | 0 | 0 | 0
  ALT >3 x ULN (n=101, 105, 97, 94) | 3 | 2 | 0 | 1
  ALT >5 x ULN (n=101, 105, 97, 94) | 1 | 1 | 0 | 0
  ALT >10 x ULN (n=101, 105, 97, 94) | 1 | 0 | 0 | 0
  ALT >20 x ULN (n=101, 105, 97, 94) | 0 | 0 | 0 | 0
  Bilirubin Total >2mg/dL (n=101, 105, 97, 94) | 1 | 0 | 3 | 0
  Bilirubin Total >1.5xULN (n=101, 105, 97, 94) | 1 | 0 | 3 | 0
  Bilirubin Total >2xULN (n=101, 105, 97, 94) | 1 | 0 | 1 | 0
  BUN >2 x pre-Rx and >ULN (n=101, 105, 97, 94) | 1 | 3 | 1 | 0
  Creatinine >2.5 mg/dL (n=101, 105, 97, 94) | 1 | 0 | 0 | 0
  Glucose, Serum Fasting < 50 mg/dL (n=0, 0, 0, 0) | 0 | 0 | 0 | 0
  Glucose, Serum Fasting > 500 mg/dL (n=0, 0, 0, 0) | 0 | 0 | 0 | 0
  Glucose, Serum Unspec. < 50 mg/dL (n=0,0,0,0) | 0 | 0 | 0 | 0
  Glucose, Serum Unspec. > 500 mg/dL (n=0,0,0,0) | 0 | 0 | 0 | 0
  Glucose, Plasma Fasting<50mg/dL(n=101, 104, 96,94) | 1 | 0 | 1 | 2
  Glucose,Plasma Fasting>500mg/dL(n=101, 104, 96,94) | 0 | 0 | 0 | 0
  Glucose, Plasma Unspec.<50mg/dL(n=102, 105, 98,95) | 7 | 4 | 4 | 3
  Glucose,Plasma Unspec.>500mg/dL(n=102, 105, 98,95) | 0 | 1 | 0 | 2
  Sodium,Serum Low (see above) (n=101, 105, 97, 94) | 0 | 0 | 0 | 1
  Sodium,Serum High(see above) (n=101, 105, 97, 94) | 1 | 0 | 1 | 0
  Potassium,Serum Low(see above)(n=101, 105, 97, 94) | 0 | 0 | 0 | 0
  Potassium, Serum High(see above)(n=101,105,97,94) | 3 | 3 | 1 | 3
  Chloride < 90 mEq/L (n=101, 105, 97, 94) | 0 | 0 | 0 | 1
  Chloride > 120 mEq/L (n=101, 105, 97, 94) | 0 | 0 | 0 | 0
  Albumin < 0.9 LLN (n=101, 105, 97, 94) | 0 | 0 | 0 | 0
  Creatine Kinase > 5 x ULN (n=101, 105, 97, 94) | 2 | 4 | 1 | 4
  Uric Acid > 1.5 x ULN (n=0, 0, 0, 0) | 0 | 0 | 0 | 0
  Protein Urine, >=2-4 (n=99, 103, 94, 92) | 8 | 9 | 4 | 3
  Blood Urine, >=2-4 (n=99, 103, 94, 92) | 5 | 11 | 8 | 16
  Red Blood Cells Urine >=2-4 (n=95, 97, 89, 88) | 6 | 8 | 8 | 14
  White Blood Cells Urine >=2-4 (n=95, 97, 89, 88) | 13 | 19 | 15 | 12

15. Other Pre Specified Outcome: Baseline and Changes From Baseline in Hemoglobin During the ST + LT Period
Time Frame: Weeks 0, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167, 180, 193, 206
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: g/dL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
g/dL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 14.49 (0.133) | 14.45 (0.125) | 14.47 (0.137) | 14.50 (0.131)
  Change from BL at Week 2 (n=95,100, 93, 87) | -0.21 (0.069) | -0.13 (0.065) | -0.22 (0.075) | -0.09 (0.078)
  Change from BL at Week 4 (n=92, 99, 91, 91) | -0.16 (0.071) | -0.15 (0.082) | -0.09 (0.069) | 0.10 (0.063)
  Change from BL at Week 6 (n=91, 96, 87, 82) | -0.12 (0.069) | -0.00 (0.074) | -0.07 (0.073) | 0.04 (0.069)
  Change from BL at Week 8 (n=92, 90, 91, 79) | -0.00 (0.068) | 0.04 (0.080) | -0.02 (0.071) | 0.09 (0.074)
  Change from BL at Week 10 (n=70, 76, 69, 63) | 0.01 (0.082) | -0.20 (0.096) | -0.13 (0.086) | 0.04 (0.097)
  Change from BL at Week 12 (n=85, 88, 87, 82) | -0.04 (0.074) | -0.07 (0.079) | -0.07 (0.083) | 0.16 (0.075)
  Change from BL at Week 14 (n=76, 80, 81, 75) | -0.09 (0.090) | -0.05 (0.078) | -0.12 (0.085) | -0.03 (0.083)
  Change from BL at Week 16 (n=90, 91, 83, 71) | -0.10 (0.087) | 0.01 (0.078) | 0.00 (0.087) | 0.04 (0.084)
  Change from BL at Week 18 (n=78, 75, 82, 71) | -0.26 (0.083) | -0.10 (0.079) | -0.07 (0.092) | -0.03 (0.099)
  Change from BL at Week 20 (n=83, 80, 78, 72) | -0.16 (0.079) | -0.14 (0.093) | -0.25 (0.081) | -0.19 (0.086)
  Change from BL at Week 22 (n=78, 74, 76, 65) | -0.35 (0.075) | -0.23 (0.092) | -0.36 (0.087) | -0.18 (0.102)
  Change from BL at Week 24 (n=83, 82, 78, 74) | -0.37 (0.079) | -0.25 (0.080) | -0.32 (0.078) | -0.14 (0.100)
  Change from BL at Week 30 (n=77, 78, 79, 67) | -0.25 (0.081) | -0.29 (0.097) | -0.19 (0.086) | -0.18 (0.101)
  Change from BL at Week 37 (n=75, 73, 70, 62) | -0.31 (0.094) | -0.22 (0.087) | -0.06 (0.090) | -0.33 (0.093)
  Change from BL at Week 50 (n=67, 71, 71, 61) | -0.17 (0.082) | 0.06 (0.103) | -0.02 (0.107) | -0.01 (0.100)
  Change from BL at Week 63 (n=61, 66, 67, 55) | -0.18 (0.112) | -0.11 (0.096) | 0.07 (0.102) | 0.08 (0.139)
  Change from BL at Week 76 (n=51, 59, 63, 49) | -0.27 (0.125) | -0.19 (0.119) | -0.07 (0.102) | -0.10 (0.117)
  Change from BL at Week 89 (n=49, 58, 56, 42) | -0.18 (0.109) | -0.09 (0.097) | -0.04 (0.103) | -0.10 (0.109)
  Change from BL at Week 102 (n=40, 49, 51, 40) | -0.32 (0.132) | -0.00 (0.129) | -0.07 (0.121) | -0.29 (0.131)
  Change from BL at Week 115 (n=34, 43, 43, 35) | -0.41 (0.132) | -0.07 (0.137) | -0.18 (0.147) | -0.19 (0.116)
  Change from BL at Week 128 (n=30, 40, 40, 30) | -0.38 (0.125) | -0.17 (0.128) | -0.25 (0.132) | -0.33 (0.124)
  Change from BL at Week 141 (n=28, 39, 34, 28) | -0.40 (0.125) | -0.35 (0.156) | -0.15 (0.169) | -0.36 (0.104)
  Change from BL at Week 154 (n=26, 34, 31, 24) | -0.45 (0.160) | -0.37 (0.186) | -0.24 (0.166) | -0.25 (0.130)
  Change from BL at Week 167 (n=24, 33, 30, 26) | -0.51 (0.178) | -0.05 (0.161) | -0.03 (0.170) | -0.24 (0.148)
  Change from BL at Week 180 (n=21, 28, 28, 26) | -0.38 (0.178) | -0.08 (0.176) | -0.08 (0.167) | -0.61 (0.169)
  Change from BL at Week 193 (n=19, 26, 26, 23) | -0.45 (0.212) | -0.03 (0.190) | -0.16 (0.178) | -0.39 (0.175)
  Change from BL at Week 206 (n=17, 22, 24, 21) | -0.51 (0.221) | -0.07 (0.195) | 0.10 (0.124) | -0.32 (0.174)

16. Other Pre Specified Outcome: Baseline and Changes From Baseline in Hematocrit During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: percentage red blood cells
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
percentage red blood cells
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 42.5 (0.35) | 42.8 (0.35) | 42.7 (0.37) | 42.8 (0.35)
  Change from BL at Week 2 (n=95,100, 93, 87) | -0.4 (0.22) | -0.2 (0.20) | -0.7 (0.21) | -0.4 (0.23)
  Change from BL at Week 4 (n=92, 99, 91, 91) | -0.2 (0.21) | -0.2 (0.24) | -0.1 (0.22) | 0.3 (0.21)
  Change from BL at Week 6 (n=91, 96, 87, 82) | 0.1 (0.19) | 0.3 (0.24) | 0.0 (0.24) | 0.3 (0.25)
  Change from BL at Week 8 (n=92, 90, 91, 79) | 0.5 (0.22) | 0.4 (0.27) | 0.2 (0.20) | 0.5 (0.25)
  Change from BL at Week 10 (n=70, 76, 69, 63) | 0.6 (0.25) | -0.0 (0.31) | -0.2 (0.24) | 0.5 (0.32)
  Change from BL at Week 12 (n=85, 88, 87, 82) | 0.6 (0.25) | 0.4 (0.26) | 0.6 (0.26) | 0.7 (0.25)
  Change from BL at Week 14 (n=76, 80, 81, 75) | 0.6 (0.27) | 0.6 (0.27) | 0.2 (0.27) | 0.2 (0.26)
  Change from BL at Week 16 (n=90. 91, 83, 71) | 0.5 (0.24) | 0.7 (0.26) | 0.6 (0.25) | 0.3 (0.30)
  Change from BL at Week 18 (n=78, 75, 82, 71) | 0.2 (0.27) | 0.4 (0.29) | 0.3 (0.24) | 0.4 (0.30)
  Change from BL at Week 20 (n=83, 80, 78, 72) | 0.7 (0.25) | 0.4 (0.31) | 0.1 (0.26) | 0.2 (0.27)
  Change from BL at Week 22 (n=78, 74, 76, 65) | 0.3 (0.27) | 0.2 (0.32) | -0.3 (0.26) | 0.5 (0.32)
  Change from BL at Week 24 (n=83, 82, 78, 74) | 0.0 (0.24) | 0.2 (0.28) | -0.1 (0.24) | 0.5 (0.32)
  Change from BL at Week 30 (n=77, 78, 79, 67) | 0.5 (0.30) | -0.1 (0.36) | 0.2 (0.30) | 0.4 (0.35)
  Change from BL at Week 37 (n=75, 73, 70, 62) | 0.0 (0.30) | -0.1 (0.27) | 0.4 (0.29) | -0.4 (0.33)
  Change from BL at Week 50 (n=67, 71, 71, 61) | 0.1 (0.29) | 0.3 (0.33) | 0.1 (0.34) | 0.2 (0.27)
  Change from BL at Week 63 (n=61, 66, 67, 55) | 0.3 (0.34) | 0.1 (0.31) | 0.6 (0.34) | 0.7 (0.43)
  Change from BL at Week 76 (n=51, 59, 63, 49) | 0.7 (0.39) | 0.5 (0.40) | 0.7 (0.35) | 0.8 (0.34)
  Change from BL at Week 89 (n=49, 58, 56, 42) | 0.9 (0.37) | 0.9 (0.34) | 1.2 (0.35) | 0.4 (0.36)
  Change from BL at Week 102 (n=40, 49, 51, 40) | -0.2 (0.37) | 0.5 (0.40) | -0.0 (0.34) | -0.7 (0.36)
  Change from BL at Week 115 (n=34, 43, 43, 35) | -0.0 (0.42) | 0.6 (0.42) | 0.2 (0.46) | 0.2 (0.40)
  Change from BL at Week 128 (n=30, 40, 40, 30) | 0.2 (0.42) | 0.3 (0.43) | 0.0 (0.43) | -0.1 (0.42)
  Change from BL at Week 141 (n=28, 39, 34, 28) | -0.1 (0.42) | -0.1 (0.48) | 0.2 (0.50) | -0.2 (0.41)
  Change from BL at Week 154 (n=26, 34, 31, 24) | -0.8 (0.45) | -0.8 (0.43) | -1.0 (0.51) | -0.3 (0.43)
  Change from BL at Week 167 (n=24, 33, 30, 26) | -0.1 (0.53) | 0.2 (0.46) | 0.2 (0.56) | -0.4 (0.48)
  Change from BL at Week 180 (n=21, 28, 28, 26) | 1.1 (0.55) | 0.6 (0.58) | 1.0 (0.53) | -0.5 (0.57)
  Change from BL at Week 193 (n=19, 26, 26, 23) | 0.6 (0.65) | 1.1 (0.55) | 0.5 (0.61) | -0.0 (0.59)
  Change from BL at Week 206 (n=17, 22, 24, 21) | -0.4 (0.54) | 0.2 (0.52) | 0.2 (0.42) | -0.5 (0.52)

17. Other Pre Specified Outcome: Baseline and Changes From Baseline in Red Blood Cell Counts (x 10^6 c/µL) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^6 c/µL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^6 c/µL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 4.80 (0.038) | 4.80 (0.042) | 4.82 (0.039) | 4.82 (0.043)
  Change from BL at Week 2 (n=95,100, 93, 87 | -0.06 (0.021) | -0.04 (0.021) | -0.08 (0.023) | -0.05 (0.023)
  Change from BL at Week 4 (n=92, 99, 91, 91) | -0.01 (0.023) | -0.04 (0.026) | -0.02 (0.022) | 0.04 (0.020)
  Change from BL at Week 6 (n=91, 96, 87, 82) | 0.00 (0.022) | 0.02 (0.024) | 0.00 (0.026) | 0.02 (0.023)
  Change from BL at Week 8 (n=92, 90, 91, 79) | 0.05 (0.020) | 0.03 (0.026) | 0.03 (0.023) | 0.05 (0.023)
  Change from BL at Week 10 (n=70, 76, 69, 63) | 0.05 (0.026) | -0.03 (0.033) | -0.02 (0.026) | 0.07 (0.032)
  Change from BL at Week 12 (n=85, 88, 87, 82) | 0.05 (0.025) | 0.03 (0.029) | 0.07 (0.025) | 0.08 (0.026)
  Change from BL at Week 14 (n=76, 80, 81, 75) | 0.05 (0.027) | 0.03 (0.029) | 0.04 (0.030) | 0.04 (0.025)
  Change from BL at Week 16 (n=90, 91, 83, 71) | 0.06 (0.027) | 0.08 (0.028) | 0.08 (0.027) | 0.06 (0.028)
  Change from BL at Week 18 (n=78, 75, 82, 71) | 0.01 (0.024) | 0.04 (0.029) | 0.05 (0.028) | 0.04 (0.030)
  Change from BL at Week 20 (n=83, 80, 78, 72) | 0.03 (0.023) | 0.02 (0.031) | 0.01 (0.025) | -0.01 (0.026)
  Change from BL at Week 22 (n=78, 74, 76, 65) | -0.01 (0.023) | -0.01 (0.033) | -0.05 (0.029) | -0.01 (0.032)
  Change from BL at Week 24 (n=83, 82, 78, 74) | -0.04 (0.024) | -0.04 (0.029) | -0.03 (0.026) | -0.01 (0.031)
  Change from BL at Week 30 (n=77, 78, 79, 67) | 0.00 (0.027) | -0.07 (0.035) | -0.01 (0.031) | -0.03 (0.034)
  Change from BL at Week 37 (n=75, 73, 70, 62) | -0.04 (0.028) | -0.04 (0.027) | 0.04 (0.031) | -0.09 (0.033)
  Change from BL at Week 50 (n=67, 71, 71, 61) | -0.02 (0.027) | 0.04 (0.031) | 0.02 (0.034) | 0.01 (0.026)
  Change from BL at Week 63 (n=61, 66, 67, 55) | 0.00 (0.032) | -0.01 (0.028) | 0.08 (0.034) | 0.05 (0.045)
  Change from BL at Week 76 (n=51, 59, 63, 49) | -0.07 (0.037) | -0.07 (0.038) | 0.00 (0.036) | -0.03 (0.037)
  Change from BL at Week 89 (n=49, 58, 56, 42) | -0.04 (0.034) | -0.06 (0.028) | -0.01 (0.035) | -0.07 (0.031)
  Change from BL at Week 102 (n=40, 49, 51, 40) | -0.10 (0.040) | -0.03 (0.043) | -0.03 (0.037) | -0.13 (0.037)
  Change from BL at Week 115 (n=34, 43, 43, 35) | -0.04 (0.039) | -0.01 (0.043) | -0.02 (0.044) | -0.06 (0.033)
  Change from BL at Week 128 (n=30, 40, 40, 30) | -0.05 (0.037) | -0.07 (0.039) | -0.04 (0.048) | -0.10 (0.039)
  Change from BL at Week 141 (n=28, 39, 34, 28) | -0.10 (0.037) | -0.13 (0.048) | -0.02 (0.052) | -0.11 (0.041)
  Change from BL at Week 154 (n=26, 35, 31, 24) | -0.13 (0.037) | -0.13 (0.045) | -0.08 (0.054) | -0.09 (0.045)
  Change from BL at Week 167 (n=24, 33, 30, 26) | -0.11 (0.052) | -0.04 (0.049) | -0.01 (0.057) | -0.10 (0.044)
  Change from BL at Week 180 (n=21, 28, 28, 26) | -0.05 (0.041) | -0.08 (0.059) | -0.01 (0.054) | -0.17 (0.056)
  Change from BL at Week 193 (n=19, 26, 26, 23) | -0.05 (0.054) | -0.06 (0.061) | -0.02 (0.057) | -0.10 (0.062)
  Change from BL at Week 206 (n=17, 22, 24, 21) | -0.03 (0.064) | -0.06 (0.058) | 0.06 (0.043) | -0.08 (0.055)

18. Other Pre Specified Outcome: Baseline and Changes From Baseline in Platelet Counts (x 10^9 c/L) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^9 c/L
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^9 c/L
  Baseline (BL) (Week 0) (n=101, 106, 96, 94) | 251.1 (6.33) | 253.1 (5.93) | 261.6 (6.71) | 259.8 (6.25)
  Change from BL at Week 2 (n=92, 96, 85, 82) | 1.8 (3.40) | 4.4 (2.82) | 2.2 (3.72) | 9.5 (3.47)
  Change from BL at Week 4 (n=88, 97, 90, 90) | 11.2 (3.39) | 8.6 (3.41) | 5.6 (3.11) | 11.3 (2.94)
  Change from BL at Week 6 (n=88, 93, 84, 81) | 4.3 (2.85) | 4.3 (3.53) | -0.2 (3.39) | 9.5 (3.05)
  Change from BL at Week 8 (n=86, 85, 86, 77) | 0.4 (3.21) | 1.0 (3.13) | -4.3 (2.94) | 4.0 (4.26)
  Change from BL at Week 10 (n=68, 75, 67, 62) | -0.8 (3.87) | 3.0 (3.99) | -4.4 (4.44) | 7.1 (3.53)
  Change from BL at Week 12 (n=83, 84, 85, 82) | -6.3 (3.58) | -1.3 (3.85) | -4.8 (4.14) | 4.0 (3.21)
  Change from BL at Week 14 (n=72, 79, 77, 74) | 1.2 (3.91) | 3.2 (4.75) | -3.7 (4.21) | 5.2 (3.59)
  Change from BL at Week 16 (n=86, 88, 81, 69) | -2.3 (3.73) | 1.1 (3.66) | -6.0 (3.74) | 3.2 (3.72)
  Change from BL at Week 18 (n=77, 71, 79, 70) | -1.1 (3.93) | 2.0 (4.06) | -2.7 (3.63) | 5.8 (3.79)
  Change from BL at Week 20 (n=78, 78, 72, 70) | -1.9 (3.87) | -4.8 (4.39) | -8.3 (3.94) | -1.3 (3.38)
  Change from BL at Week 22 (n=74, 72, 73, 62) | 0.3 (4.64) | -2.5 (3.91) | -5.4 (4.01) | 5.0 (3.48)
  Change from BL at Week 24 (n=80, 76, 73, 72) | -7.1 (3.94) | -6.0 (4.00) | -15.5 (4.54) | -3.0 (3.66)
  Change from BL at Week 30 (n=73, 74, 74, 67) | -2.0 (5.66) | -3.3 (4.37) | -9.9 (4.34) | 4.5 (4.08)
  Change from BL at Week 37 (n=70, 68, 66, 59) | -14.3 (3.85) | -8.1 (4.71) | -15.6 (3.93) | 0.1 (4.81)
  Change from BL at Week 50 (n=66, 67, 66, 59) | -2.5 (4.25) | -5.6 (4.39) | -11.5 (3.76) | 6.6 (6.29)
  Change from BL at Week 63 (n=59, 64, 65, 54) | -3.1 (4.57) | -3.4 (4.24) | -6.3 (4.23) | 10.2 (5.37)
  Change from BL at Week 76 (n=50, 58, 61, 49) | -2.0 (5.64) | -1.5 (4.56) | -6.0 (3.68) | 1.2 (4.88)
  Change from BL at Week 89 (n=47, 56, 54, 42) | 3.5 (5.29) | 1.9 (5.02) | -6.7 (3.83) | 2.7 (4.97)
  Change from BL at Week 102 (n=39, 47, 49, 39) | 3.2 (7.75) | -2.3 (5.34) | -4.8 (3.65) | 9.7 (7.21)
  Change from BL at Week 115 (n=33, 41, 41, 34) | 5.0 (8.04) | -8.8 (4.96) | -12.0 (4.23) | 9.2 (7.57)
  Change from BL at Week 128 (n=30, 38, 39, 30) | 3.8 (5.74) | -2.1 (5.39) | -2.6 (5.04) | 2.6 (7.91)
  Change from BL at Week 141 (n=27, 39, 33, 27) | -1.1 (5.34) | -4.6 (5.16) | -0.3 (4.73) | -1.3 (8.24)
  Change from BL at Week 154 (n=25, 35, 31, 23) | 5.0 (6.95) | 5.8 (7.20) | -2.9 (5.25) | 8.8 (13.59)
  Change from BL at Week 167 (n=22, 32, 28, 26) | -18.0 (6.71) | -0.1 (6.99) | -14.6 (6.21) | 4.3 (8.63)
  Change from BL at Week 180 (n=20, 27, 27, 25) | -11.1 (6.57) | -24.0 (6.18) | -17.3 (6.54) | 4.0 (10.72)
  Change from BL at Week 193 (n=17, 25, 25, 22) | -13.6 (8.11) | -13.4 (9.58) | -13.4 (6.00) | -12.0 (7.27)
  Change from BL at Week 206 (n=15, 21, 23, 21) | -2.6 (10.45) | -18.7 (9.01) | 6.2 (9.35) | -6.1 (11.49)

19. Other Pre Specified Outcome: Baseline and Changes From Baseline in White Blood Cell Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^3 c/µL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 6.71 (0.179) | 6.75 (0.198) | 6.82 (0.155) | 6.79 (0.182)
  Change from BL at Week 2 (n=95, 99, 92, 86) | -0.11 (0.136) | 0.05 (0.132) | -0.14 (0.113) | -0.23 (0.156)
  Change from BL at Week 4 (n=92, 99, 90, 90) | 0.06 (0.132) | 0.05 (0.125) | -0.16 (0.132) | 0.17 (0.137)
  Change from BL at Week 6 (n=89, 95, 87, 82) | 0.01 (0.115) | 0.10 (0.126) | -0.18 (0.128) | 0.09 (0.172)
  Change from BL at Week 8 (n=91, 89, 90, 79) | -0.02 (0.132) | 0.18 (0.144) | -0.17 (0.121) | 0.16 (0.149)
  Change from BL at Week 10 (n=68, 76, 69, 63) | 0.32 (0.168) | 0.55 (0.169) | 0.12 (0.162) | 0.53 (0.208)
  Change from BL at Week 12 (n=83, 88, 87, 82) | -0.00 (0.148) | 0.09 (0.155) | 0.05 (0.145) | 0.26 (0.163)
  Change from BL at Week 14 (n=76, 78, 80, 75) | 0.33 (0.196) | 0.71 (0.166) | 0.22 (0.134) | 0.56 (0.192)
  Change from BL at Week 16 (n=90, 91, 83, 71) | 0.24 (0.146) | 0.54 (0.148) | 0.04 (0.138) | 0.19 (0.163)
  Change from BL at Week 18 (n=78, 75, 82, 71) | 0.37 (0.166) | 0.82 (0.172) | 0.42 (0.142) | 0.32 (0.185)
  Change from BL at Week 20 (n=83, 79, 78, 72) | 0.29 (0.150) | 0.29 (0.163) | 0.01 (0.140) | 0.02 (0.154)
  Change from BL at Week 22 (n=77, 74, 76, 65) | 0.66 (0.184) | 0.72 (0.178) | 0.44 (0.175) | 0.45 (0.163)
  Change from BL at Week 24 (n=83, 82, 78, 74) | 0.10 (0.149) | 0.47 (0.265) | 0.08 (0.158) | -0.06 (0.142)
  Change from BL at Week 30 (n=77, 78, 79, 67) | 0.15 (0.148) | 0.33 (0.202) | 0.28 (0.167) | -0.03 (0.129)
  Change from BL at Week 37 (n=74, 73, 70, 62) | 0.21 (0.163) | 0.42 (0.204) | 0.12 (0.189) | 0.14 (0.159)
  Change from BL at Week 50 (n=67, 69, 71, 61) | 0.01 (0.168) | 0.33 (0.216) | -0.03 (0.149) | 0.29 (0.186)
  Change from BL at Week 63 (n=60, 66, 67, 55) | 0.12 (0.176) | 0.20 (0.221) | -0.04 (0.180) | 0.06 (0.176)
  Change from BL at Week 76 (n=51, 58, 63, 49) | 0.03 (0.185) | 0.23 (0.259) | -0.07 (0.158) | -0.20 (0.169)
  Change from BL at Week 89 (n=48, 58, 56, 42) | 0.51 (0.232) | 0.17 (0.246) | -0.10 (0.152) | -0.18 (0.232)
  Change from BL at Week 102 (n=39, 47, 51, 40) | 0.16 (0.218) | 0.44 (0.258) | 0.10 (0.129) | -0.09 (0.208)
  Change from BL at Week 115 (n=34, 43, 42, 34) | 0.24 (0.235) | 0.93 (0.252) | 0.11 (0.210) | 0.44 (0.286)
  Change from BL at Week 128 (n=30, 40, 40, 29) | 0.58 (0.227) | 0.66 (0.314) | 0.44 (0.221) | 0.22 (0.286)
  Change from BL at Week 141 (n=28, 39, 34, 28) | 0.35 (0.183) | 0.78 (0.303) | 0.44 (0.199) | 0.51 (0.214)
  Change from BL at Week 154 (n=26, 34, 31, 24) | 0.12 (0.228) | 0.44 (0.327) | 0.30 (0.212) | 0.38 (0.217)
  Change from BL at Week 167 (n=24, 33, 30, 25) | -0.22 (0.233) | 0.44 (0.341) | 0.27 (0.209) | 0.35 (0.180)
  Change from BL at Week 180 (n=21, 28, 28, 26) | 0.13 (0.233) | 0.30 (0.379) | 0.59 (0.263) | 0.65 (0.267)
  Change from BL at Week 193 (n=19, 26, 26, 23) | 0.34 (0.220) | 0.02 (0.403) | 0.60 (0.205) | 0.19 (0.157)
  Change from BL at Week 206 (n=17, 22, 23, 21) | 0.01 (0.199) | 0.55 (0.420) | 1.01 (0.303) | 0.38 (0.284)

20. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Neutrophil Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^3 c/µL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 4.00 (0.141) | 3.98 (0.142) | 4.16 (0.137) | 4.01 (0.148)
  Change from BL at Week 2 (n=95, 99, 92, 86) | -0.06 (0.122) | 0.11 (0.117) | 0.00 (0.101) | -0.07 (0.131)
  Change from BL at Week 4 (n=91, 99, 90, 90) | 0.09 (0.114) | 0.16 (0.103) | 0.05 (0.121) | 0.23 (0.120)
  Change from BL at Week 6 (n=89, 95, 87, 82) | 0.01 (0.105) | 0.19 (0.097) | 0.04 (0.114) | 0.17 (0.150)
  Change from BL at Week 8 (n=91, 88, 90, 79) | 0.02 (0.110) | 0.27 (0.131) | 0.03 (0.096) | 0.19 (0.126)
  Change from BL at Week 10 (n=68, 76, 69, 63) | 0.18 (0.135) | 0.48 (0.145) | 0.17 (0.139) | 0.45 (0.169)
  Change from BL at Week 12 (n=83, 88, 87, 82) | 0.01 (0.135) | 0.21 (0.130) | 0.18 (0.115) | 0.30 (0.139)
  Change from BL at Week 14 (n=76, 77, 80, 75) | 0.07 (0.158) | 0.64 (0.119) | 0.17 (0.115) | 0.46 (0.161)
  Change from BL at Week 16 (n=90, 91, 83, 71) | 0.17 (0.116) | 0.49 (0.132) | 0.16 (0.132) | 0.18 (0.140)
  Change from BL at Week 18 (n=78, 75, 82, 71) | 0.23 (0.120) | 0.67 (0.149) | 0.32 (0.130) | 0.21 (0.148)
  Change from BL at Week 20 (n=83, 79, 78, 72) | 0.19 (0.131) | 0.32 (0.141) | 0.07 (0.130) | 0.15 (0.127)
  Change from BL at Week 22 (n=77, 74, 75, 65) | 0.44 (0.155) | 0.58 (0.160) | 0.44 (0.153) | 0.32 (0.130)
  Change from BL at Week 24 (n=83, 81, 78, 74) | 0.09 (0.124) | 0.57 (0.263) | 0.16 (0.130) | -0.03 (0.115)
  Change from BL at Week 30 (n=76, 78, 79, 67) | 0.04 (0.124) | 0.29 (0.155) | 0.32 (0.122) | 0.00 (0.114)
  Change from BL at Week 37 (n=74, 72, 70, 60) | 0.13 (0.146) | 0.42 (0.171) | 0.24 (0.165) | 0.20 (0.137)
  Change from BL at Week 50 (n=67, 69, 71, 61) | 0.03 (0.144) | 0.40 (0.182) | 0.19 (0.128) | 0.27 (0.161)
  Change from BL at Week 63 (n=60, 66, 67, 55) | 0.11 (0.140) | 0.25 (0.176) | 0.08 (0.168) | 0.16 (0.152)
  Change from BL at Week 76 (n=51, 58, 63, 49) | 0.05 (0.161) | 0.33 (0.204) | 0.08 (0.146) | -0.01 (0.140)
  Change from BL at Week 89 (n=48, 58, 56, 42) | 0.58 (0.208) | 0.18 (0.178) | 0.05 (0.136) | 0.01 (0.185)
  Change from BL at Week 102 (n=39, 47, 50, 40) | 0.19 (0.212) | 0.43 (0.215) | 0.24 (0.114) | 0.01 (0.176)
  Change from BL at Week 115 (n=34, 43, 42, 34) | 0.28 (0.219) | 0.81 (0.165) | 0.29 (0.178) | 0.42 (0.223)
  Change from BL at Week 128 (n=30, 40, 40, 29) | 0.61 (0.202) | 0.59 (0.244) | 0.56 (0.209) | 0.22 (0.245)
  Change from BL at Week 141 (n=28, 38, 34, 28) | 0.41 (0.168) | 0.80 (0.254) | 0.45 (0.161) | 0.40 (0.198)
  Change from BL at Week 154 (n=26, 33, 31, 24) | 0.25 (0.223) | 0.39 (0.225) | 0.47 (0.162) | 0.41 (0.184)
  Change from BL at Week 167 (n=24, 33, 30, 25) | -0.04 (0.211) | 0.56 (0.239) | 0.27 (0.193) | 0.33 (0.176)
  Change from BL at Week 180 (n=21, 28, 28, 26) | 0.23 (0.220) | 0.50 (0.293) | 0.55 (0.200) | 0.51 (0.271)
  Change from BL at Week 193 (n=19, 25, 26, 23) | 0.34 (0.181) | 0.08 (0.277) | 0.51 (0.166) | -0.01 (0.130)
  Change from BL at Week 206 (n=17, 22, 23, 21) | 0.15 (0.218) | 0.63 (0.389) | 0.90 (0.284) | 0.31 (0.235)

21. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Lymphocyte Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^3 c/µL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 2.16 (0.062) | 2.21 (0.071) | 2.14 (0.063) | 2.22 (0.063)
  Change from BL at Week 2 (n=95, 99, 92, 86) | -0.04 (0.052) | -0.10 (0.045) | -0.11 (0.046) | -0.13 (0.049)
  Change from BL at Week 4 (n=91, 99, 90, 90) | -0.03 (0.056) | -0.12 (0.046) | -0.18 (0.046) | -0.04 (0.040)
  Change from BL at Week 6 (n=89, 95, 87, 82) | -0.04 (0.049) | -0.09 (0.057) | -0.23 (0.047) | -0.09 (0.048)
  Change from BL at Week 8 (n=91, 88, 90, 79) | -0.07 (0.049) | -0.11 (0.049) | -0.20 (0.048) | -0.00 (0.053)
  Change from BL at Week 10 (n=68, 76, 69, 63) | 0.07 (0.069) | 0.02 (0.055) | -0.10 (0.053) | 0.05 (0.068)
  Change from BL at Week 12 (n=83, 88, 87, 82) | -0.06 (0.049) | -0.12 (0.044) | -0.16 (0.052) | -0.02 (0.058)
  Change from BL at Week 14 (n=76, 77, 80, 75) | 0.20 (0.071) | 0.08 (0.085) | -0.01 (0.052) | 0.06 (0.058)
  Change from BL at Week 16 (n=90, 91, 83, 71) | 0.03 (0.065) | 0.01 (0.057) | -0.11 (0.049) | 0.01 (0.061)
  Change from BL at Week 18 (n=78, 75, 82, 71) | 0.11 (0.079) | 0.13 (0.064) | 0.01 (0.064) | 0.08 (0.069)
  Change from BL at Week 20 (n=83, 79, 78, 72) | 0.08 (0.065) | -0.02 (0.064) | -0.10 (0.058) | -0.11 (0.052)
  Change from BL at Week 22 (n=77, 74, 75, 65) | 0.16 (0.069) | 0.13 (0.083) | -0.07 (0.060) | 0.09 (0.067)
  Change from BL at Week 24 (n=83, 81, 78, 74) | -0.00 (0.068) | -0.07 (0.071) | -0.13 (0.054) | -0.01 (0.059)
  Change from BL at Week 30 (n=76, 78, 79, 67) | 0.08 (0.066) | -0.00 (0.060) | -0.09 (0.063) | -0.03 (0.059)
  Change from BL at Week 37 (n=74, 72, 70, 60) | 0.05 (0.067) | 0.02 (0.064) | -0.17 (0.056) | -0.08 (0.066)
  Change from BL at Week 50 (n=67, 69, 71, 61) | -0.06 (0.071) | -0.09 (0.069) | -0.25 (0.051) | -0.03 (0.059)
  Change from BL at Week 63 (n=60, 66, 67, 55) | -0.06 (0.077) | -0.10 (0.063) | -0.19 (0.070) | -0.16 (0.063)
  Change from BL at Week 76 (n=51, 58, 63, 49) | -0.10 (0.086) | -0.09 (0.082) | -0.18 (0.054) | -0.20 (0.072)
  Change from BL at Week 89 (n=49, 58, 56, 42) | -0.12 (0.087) | -0.02 (0.080) | -0.19 (0.054) | -0.23 (0.083)
  Change from BL at Week 102 (n=39, 48, 51, 40) | -0.17 (0.081) | -0.07 (0.086) | -0.23 (0.056) | -0.16 (0.071)
  Change from BL at Week 115 (n=34, 43, 43, 35) | -0.15 (0.080) | -0.00 (0.103) | -0.21 (0.068) | -0.10 (0.100)
  Change from BL at Week 128 (n=30, 40, 40, 30) | -0.12 (0.106) | -0.00 (0.105) | -0.16 (0.068) | -0.06 (0.094)
  Change from BL at Week 141 (n=28, 38, 34, 28) | -0.13 (0.089) | -0.03 (0.083) | -0.10 (0.079) | 0.00 (0.086)
  Change from BL at Week 154 (n=26, 33, 31, 24) | -0.23 (0.096) | 0.04 (0.128) | -0.23 (0.101) | -0.14 (0.096)
  Change from BL at Week 167 (n=24, 33, 30, 25) | -0.23 (0.096) | -0.13 (0.118) | -0.11 (0.090) | -0.16 (0.084)
  Change from BL at Week 180 (n=21, 28, 28, 26) | -0.15 (0.107) | -0.22 (0.130) | -0.06 (0.105) | -0.05 (0.102)
  Change from BL at Week 193 (n=19, 25, 26, 23) | -0.06 (0.094) | -0.09 (0.151) | -0.04 (0.092) | 0.01 (0.101)
  Change from BL at Week 206 (n=17, 22, 23, 21) | -0.17 (0.126) | -0.14 (0.105) | -0.05 (0.094) | -0.08 (0.113)

22. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Monocyte Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^3 c/µL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 0.31 (0.016) | 0.34 (0.017) | 0.32 (0.016) | 0.32 (0.015)
  Change from BL at Week 2 (n=95, 99, 92, 86) | 0.01 (0.015) | 0.01 (0.017) | -0.05 (0.021) | -0.01 (0.018)
  Change from BL at Week 4 (n=91, 99, 90, 90) | 0.05 (0.015) | 0.00 (0.014) | -0.01 (0.020) | 0.01 (0.015)
  Change from BL at Week 6 (n=89, 95, 87, 82) | 0.05 (0.017) | -0.01 (0.017) | -0.01 (0.019) | 0.02 (0.019)
  Change from BL at Week 8 (n=91, 88, 90, 79) | 0.03 (0.016) | 0.03 (0.018) | -0.01 (0.017) | -0.02 (0.018)
  Change from BL at Week 10 (n=68, 76, 69, 63) | 0.08 (0.020) | 0.04 (0.021) | 0.04 (0.021) | 0.03 (0.024)
  Change from BL at Week 12 (n=83, 88, 87, 82) | 0.05 (0.017) | 0.00 (0.018) | 0.00 (0.019) | 0.01 (0.018)
  Change from BL at Week 14 (n=76, 77, 80, 75) | 0.09 (0.019) | 0.06 (0.022) | 0.03 (0.021) | 0.04 (0.021)
  Change from BL at Week 16 (n=90, 91, 83, 71) | 0.06 (0.018) | 0.04 (0.019) | 0.04 (0.019) | 0.01 (0.017)
  Change from BL at Week 18 (n=78, 75, 82, 71) | 0.06 (0.018) | 0.05 (0.025) | 0.06 (0.018) | 0.04 (0.021)
  Change from BL at Week 20 (n=83, 79, 78, 72) | 0.04 (0.017) | 0.02 (0.018) | 0.04 (0.021) | 0.01 (0.022)
  Change from BL at Week 22 (n=77, 74, 75, 65) | 0.08 (0.023) | 0.05 (0.017) | 0.06 (0.021) | 0.05 (0.021)
  Change from BL at Week 24 (n=83, 81, 78, 74) | 0.04 (0.019) | 0.01 (0.019) | 0.03 (0.019) | 0.03 (0.019)
  Change from BL at Week 30 (n=76, 78, 79, 67) | 0.05 (0.020) | 0.03 (0.022) | 0.04 (0.021) | 0.03 (0.018)
  Change from BL at Week 37 (n=74, 72, 70, 60) | 0.06 (0.022) | 0.02 (0.022) | 0.04 (0.020) | 0.00 (0.020)
  Change from BL at Week 50 (n=67, 69, 71, 61) | 0.07 (0.021) | 0.03 (0.020) | 0.05 (0.022) | 0.06 (0.018)
  Change from BL at Week 63 (n=60, 66, 67, 55) | 0.08 (0.021) | 0.05 (0.022) | 0.07 (0.026) | 0.07 (0.019)
  Change from BL at Week 76 (n=51, 58, 63, 49) | 0.12 (0.026) | 0.04 (0.028) | 0.06 (0.024) | 0.05 (0.020)
  Change from BL at Week 89 (n=48, 58, 56, 42) | 0.11 (0.023) | 0.03 (0.026) | 0.08 (0.022) | 0.05 (0.028)
  Change from BL at Week 102 (n=39, 47, 50, 40) | 0.14 (0.025) | 0.04 (0.028) | 0.09 (0.028) | 0.07 (0.025)
  Change from BL at Week 115 (n=34, 43, 42, 34) | 0.12 (0.033) | 0.05 (0.026) | 0.06 (0.029) | 0.13 (0.030)
  Change from BL at Week 128 (n=30, 40, 40, 29) | 0.12 (0.031) | 0.04 (0.031) | 0.07 (0.026) | 0.07 (0.022)
  Change from BL at Week 141 (n=28, 38, 34, 28) | 0.08 (0.029) | 0.02 (0.030) | 0.10 (0.028) | 0.10 (0.024)
  Change from BL at Week 154 (n=26, 33, 31, 24) | 0.10 (0.025) | 0.05 (0.037) | 0.06 (0.035) | 0.08 (0.022)
  Change from BL at Week 167 (n=24, 33, 30, 25) | 0.07 (0.029) | 0.04 (0.036) | 0.10 (0.036) | 0.11 (0.023)
  Change from BL at Week 180 (n=21, 28, 28, 26) | 0.08 (0.028) | 0.04 (0.041) | 0.11 (0.040) | 0.11 (0.021)
  Change from BL at Week 193 (n=19, 25, 26, 23) | 0.09 (0.039) | 0.04 (0.044) | 0.11 (0.036) | 0.13 (0.023)
  Change from BL at Week 206 (n=17, 22, 23, 21) | 0.05 (0.033) | 0.05 (0.034) | 0.13 (0.042) | 0.09 (0.023)

23. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Basophil Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^3 c/µL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 0.01 (0.003) | 0.02 (0.004) | 0.02 (0.004) | 0.02 (0.004)
  Change from BL at Week 2 (n=95, 99, 92, 86) | 0.00 (0.004) | -0.01 (0.004) | -0.01 (0.004) | 0.00 (0.005)
  Change from BL at Week 4 (n=91, 99, 90, 90) | 0.00 (0.004) | -0.01 (0.004) | -0.01 (0.003) | -0.00 (0.005)
  Change from BL at Week 6 (n=89, 95, 87, 82) | 0.01 (0.005) | -0.01 (0.004) | -0.01 (0.004) | -0.01 (0.005)
  Change from BL at Week 8 (n=91, 88, 90, 79) | 0.00 (0.003) | -0.00 (0.005) | -0.01 (0.004) | -0.01 (0.005)
  Change from BL at Week 10 (n=68, 76, 69, 63) | 0.00 (0.004) | -0.01 (0.004) | -0.01 (0.004) | -0.01 (0.005)
  Change from BL at Week 12 (n=83, 88, 87, 82) | -0.00 (0.004) | -0.01 (0.005) | -0.00 (0.004) | -0.00 (0.005)
  Change from BL at Week 14 (n=76, 77, 80, 75) | 0.00 (0.004) | 0.00 (0.006) | -0.01 (0.004) | -0.00 (0.005)
  Change from BL at Week 16 (n=90, 91, 83, 71) | 0.00 (0.004) | -0.00 (0.005) | -0.01 (0.003) | -0.01 (0.006)
  Change from BL at Week 18 (n=78, 75, 82, 71) | 0.00 (0.004) | 0.00 (0.005) | -0.00 (0.006) | -0.01 (0.005)
  Change from BL at Week 20 (n=83, 79, 78, 72) | 0.01 (0.004) | -0.01 (0.005) | -0.01 (0.004) | -0.00 (0.005)
  Change from BL at Week 22 (n=77, 74, 75, 65) | 0.01 (0.004) | -0.00 (0.005) | 0.00 (0.013) | -0.00 (0.006)
  Change from BL at Week 24 (n=83, 81, 78, 74) | 0.00 (0.005) | -0.01 (0.004) | -0.01 (0.005) | -0.01 (0.006)
  Change from BL at Week 30 (n=76, 78, 79, 67) | 0.00 (0.004) | 0.01 (0.006) | -0.01 (0.005) | 0.01 (0.006)
  Change from BL at Week 37 (n=74, 72, 70, 60) | 0.00 (0.004) | 0.01 (0.006) | 0.00 (0.005) | 0.00 (0.007)
  Change from BL at Week 50 (n=67, 69, 71, 61) | 0.02 (0.004) | 0.01 (0.006) | 0.01 (0.005) | 0.02 (0.005)
  Change from BL at Week 63 (n=60, 66, 67, 55) | 0.02 (0.005) | 0.01 (0.005) | 0.02 (0.006) | 0.02 (0.004)
  Change from BL at Week 76 (n=51, 58, 63, 49) | 0.02 (0.004) | 0.01 (0.005) | 0.02 (0.005) | 0.01 (0.005)
  Change from BL at Week 89 (n=48, 58, 56, 42) | 0.02 (0.006) | 0.02 (0.006) | 0.02 (0.005) | 0.02 (0.006)
  Change from BL at Week 102 (n=39, 47, 50, 40) | 0.02 (0.007) | 0.02 (0.005) | 0.02 (0.005) | 0.02 (0.007)
  Change from BL at Week 115 (n=34, 43, 42, 34) | 0.02 (0.006) | 0.03 (0.007) | 0.01 (0.007) | 0.03 (0.008)
  Change from BL at Week 128 (n=30, 40, 40, 29) | 0.03 (0.008) | 0.03 (0.007) | 0.01 (0.006) | 0.03 (0.008)
  Change from BL at Week 141 (n=28, 38, 34, 28) | 0.02 (0.008) | 0.02 (0.007) | 0.01 (0.007) | 0.02 (0.009)
  Change from BL at Week 154 (n=26, 33, 31, 24) | 0.03 (0.008) | 0.02 (0.006) | 0.02 (0.009) | 0.01 (0.010)
  Change from BL at Week 167 (n=24, 33, 30, 25) | 0.02 (0.009) | 0.01 (0.008) | 0.01 (0.008) | 0.02 (0.008)
  Change from BL at Week 180 (n=21, 28, 28, 26) | 0.01 (0.007) | 0.02 (0.007) | 0.00 (0.007) | 0.02 (0.009)
  Change from BL at Week 193 (n=19, 25, 26, 23) | 0.01 (0.010) | 0.01 (0.009) | 0.01 (0.008) | 0.02 (0.008)
  Change from BL at Week 206 (n=17, 22, 23, 21) | 0.00 (0.013) | 0.02 (0.010) | 0.01 (0.010) | 0.01 (0.009)

24. Other Pre Specified Outcome: Baseline and Changes From Baseline in Absolute Eosinophil Counts (x 10^3 c/µL) During the ST + LT Period
Time Frame: as for outcome 15
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: x 10^3 c/µL
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
x 10^3 c/µL
  Baseline (BL) (Week 0) (n=102, 106, 98, 94) | 0.18 (0.012) | 0.20 (0.015) | 0.20 (0.012) | 0.20 (0.016)
  Change from BL at Week 2 (n=95, 99, 92, 86) | -0.01 (0.008) | 0.01 (0.011) | -0.02 (0.009) | -0.02 (0.013)
  Change from BL at Week 4 (n=91, 99, 90, 90) | -0.02 (0.011) | -0.01 (0.012) | -0.01 (0.011) | -0.02 (0.012)
  Change from BL at Week 6 (n=89, 95, 87, 82) | 0.01 (0.009) | -0.01 (0.012) | -0.02 (0.011) | -0.02 (0.014)
  Change from BL at Week 8 (n=91, 88, 90, 79) | 0.00 (0.011) | -0.01 (0.014) | -0.02 (0.012) | -0.01 (0.015)
  Change from BL at Week 10 (n=68, 76, 69, 63) | -0.01 (0.014) | -0.02 (0.015) | -0.02 (0.013) | 0.01 (0.015)
  Change from BL at Week 12 (n=83, 88, 87, 82) | 0.00 (0.024) | -0.02 (0.014) | -0.01 (0.015) | -0.02 (0.013)
  Change from BL at Week 14 (n=76, 77, 80, 75) | -0.01 (0.015) | -0.01 (0.017) | -0.01 (0.019) | -0.01 (0.017)
  Change from BL at Week 16 (n=90, 91, 83, 71) | -0.02 (0.010) | -0.02 (0.014) | -0.03 (0.014) | -0.00 (0.018)
  Change from BL at Week 18 (n=78, 75, 82, 71) | -0.02 (0.011) | -0.02 (0.018) | -0.03 (0.013) | 0.00 (0.020)
  Change from BL at Week 20 (n=83, 79, 78, 72) | -0.02 (0.012) | -0.03 (0.015) | -0.04 (0.012) | -0.03 (0.016)
  Change from BL at Week 22 (n=77, 74, 75, 65) | -0.00 (0.015) | -0.03 (0.013) | -0.04 (0.012) | -0.02 (0.016)
  Change from BL at Week 24 (n=83, 81, 78, 74) | -0.02 (0.013) | -0.03 (0.015) | -0.03 (0.011) | -0.04 (0.016)
  Change from BL at Week 30 (n=76, 78, 79, 67) | -0.03 (0.013) | -0.03 (0.017) | -0.02 (0.011) | -0.03 (0.016)
  Change from BL at Week 37 (n=74, 72, 70, 60) | -0.03 (0.010) | -0.01 (0.019) | -0.04 (0.012) | -0.02 (0.020)
  Change from BL at Week 50 (n=67, 69, 71, 61) | -0.03 (0.013) | -0.01 (0.019) | -0.02 (0.011) | -0.01 (0.018)
  Change from BL at Week 63 (n=60, 66, 67, 55) | -0.00 (0.019) | 0.00 (0.025) | -0.00 (0.017) | -0.02 (0.013)
  Change from BL at Week 76 (n=51, 58, 63, 49) | -0.03 (0.014) | -0.04 (0.022) | -0.02 (0.013) | -0.03 (0.020)
  Change from BL at Week 89 (n=48, 58, 56, 42) | -0.03 (0.019) | -0.02 (0.025) | -0.02 (0.013) | -0.02 (0.020)
  Change from BL at Week 102 (n=39, 47, 50, 40) | 0.02 (0.025) | 0.01 (0.027) | 0.02 (0.016) | -0.01 (0.018)
  Change from BL at Week 115 (n=34, 43, 42, 34) | -0.00 (0.019) | 0.07 (0.051) | -0.01 (0.019) | -0.00 (0.023)
  Change from BL at Week 128 (n=30, 40, 40, 29) | -0.02 (0.017) | 0.02 (0.046) | -0.03 (0.014) | -0.01 (0.025)
  Change from BL at Week 141 (n=28, 38, 34, 28) | -0.01 (0.020) | -0.00 (0.019) | -0.00 (0.016) | 0.01 (0.020)
  Change from BL at Week 154 (n=26, 33, 31, 24) | 0.00 (0.017) | -0.00 (0.019) | -0.01 (0.018) | 0.03 (0.021)
  Change from BL at Week 167 (n=24, 33, 30, 25) | -0.02 (0.014) | -0.02 (0.020) | 0.01 (0.017) | 0.06 (0.039)
  Change from BL at Week 180 (n=21, 28, 28, 26) | -0.02 (0.013) | -0.01 (0.021) | -0.00 (0.014) | 0.07 (0.040)
  Change from BL at Week 193 (n=19, 25, 26, 23) | -0.01 (0.019) | -0.01 (0.024) | 0.00 (0.017) | 0.05 (0.032)
  Change from BL at Week 206 (n=17, 22, 23, 21) | 0.00 (0.026) | -0.00 (0.028) | 0.03 (0.016) | 0.06 (0.026)

25. Other Pre Specified Outcome: Changes From Baseline in Systolic Blood Pressure During the ST + LT Period
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167, 180, 193, 206
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
mmHg
  Change from BL at Week 2 (n=96, 100, 94, 89) | -1.0 (1.4) | -2.0 (1.3) | -2.3 (1.2) | -3.1 (1.4)
  Change from BL at Week 4 (n=96, 100, 92, 91) | -1.9 (1.4) | -1.2 (1.1) | -2.3 (1.1) | -4.3 (1.4)
  Change from BL at Week 6 (n=91, 98, 88, 84) | -1.5 (1.4) | -2.1 (1.2) | -3.5 (1.3) | -4.5 (1.4)
  Change from BL at Week 8 (n=94, 91, 91, 80) | -3.0 (1.4) | -1.8 (1.2) | -4.0 (1.2) | -5.5 (1.5)
  Change from BL at Week 10 (n=51, 66, 51, 50) | -3.6 (2.0) | -2.9 (1.5) | -5.0 (1.5) | -6.1 (1.7)
  Change from BL at Week 12 (n=82, 83, 87, 79) | -3.3 (1.3) | -2.9 (1.2) | -2.8 (1.3) | -3.2 (1.6)
  Change from BL at Week 14 (n=65, 72, 66, 62) | -4.9 (1.6) | -2.0 (1.5) | -6.0 (1.7) | -1.9 (1.6)
  Change from BL at Week 16 (n=87, 87, 81, 72) | -3.2 (1.4) | -2.1 (1.3) | -3.8 (1.4) | -2.1 (1.5)
  Change from BL at Week 18 (n=73, 69, 76, 66) | -5.1 (1.7) | -0.9 (1.5) | -4.3 (1.7) | -4.7 (1.9)
  Change from BL at Week 20 (n=84, 80, 76, 73) | -5.0 (1.6) | -3.2 (1.3) | -3.3 (1.4) | -4.9 (1.7)
  Change from BL at Week 22 (n=78, 73, 76, 64) | -6.1 (1.7) | -4.5 (1.3) | -5.9 (1.5) | -3.9 (1.9)
  Change from BL at Week 24 (n=84, 83, 77, 75) | -2.8 (1.5) | -4.1 (1.2) | -6.2 (1.5) | -6.3 (1.7)
  Change from BL at Week 30 (n=79, 78, 79, 66) | -3.6 (1.7) | -3.8 (1.5) | -3.9 (1.5) | -5.4 (1.9)
  Change from BL at Week 37 (n=77, 74, 71, 66) | -3.0 (1.7) | -3.5 (1.4) | -5.2 (1.5) | -3.6 (1.7)
  Change from BL at Week 50 (n=70, 73, 73, 62) | -2.5 (1.7) | 0.1 (1.4) | -3.3 (1.5) | -0.4 (1.9)
  Change from BL at Week 63 (n=62, 66, 69, 56) | -1.2 (1.9) | -0.3 (1.4) | -1.1 (1.5) | -2.4 (2.1)
  Change from BL at Week 76 (n=53, 59, 64, 50) | -2.9 (1.7) | -2.6 (1.6) | -3.1 (1.8) | -0.9 (2.2)
  Change from BL at Week 89 (n=49, 58, 56, 44) | -2.8 (2.0) | -3.4 (1.4) | -5.4 (2.0) | -2.2 (2.2)
  Change from BL at Week 102 (n=42, 47, 50, 40) | -0.6 (2.1) | -1.1 (1.9) | -2.9 (2.1) | -1.0 (2.5)
  Change from BL at Week 115 (n=34, 43, 43, 37) | -2.6 (2.4) | -2.6 (2.0) | -1.6 (1.9) | 0.9 (2.7)
  Change from BL at Week 128 (n=31, 40, 41, 31) | -5.1 (2.5) | -5.5 (1.9) | 0.0 (1.9) | 1.1 (2.7)
  Change from BL at Week 141 (n=29, 40, 35, 29) | -1.8 (3.0) | -5.2 (2.3) | 0.3 (2.6) | -1.4 (3.1)
  Change from BL at Week 154 (n=27, 36, 33, 27) | -0.8 (2.8) | -0.5 (2.3) | 3.5 (2.6) | 2.3 (3.1)
  Change from BL at Week 167 (n=24, 33, 30, 27) | 0.7 (2.9) | -1.8 (2.5) | 4.0 (2.5) | -0.6 (3.1)
  Change from BL at Week 180 (n=21, 28, 28, 27) | 0.9 (2.9) | -5.4 (3.2) | 0.9 (2.4) | -0.8 (2.6)
  Change from BL at Week 193 (n=19, 26, 27, 24) | 3.4 (4.0) | -7.5 (3.2) | 0.0 (3.0) | -2.6 (3.6)
  Change from BL at Week 206 (n=17, 24, 24, 23) | 4.8 (5.0) | -2.8 (3.3) | 2.3 (2.6) | 0.7 (4.0)

26. Other Pre Specified Outcome: Changes From Baseline in Diastolic Blood Pressure During the ST + LT Period
Time Frame: as for outcome 25
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
mmHg
  Change from BL at Week 2 (n=96, 100, 94, 89) | -0.0 (0.7) | -1.2 (0.8) | -0.5 (0.7) | -1.5 (0.9)
  Change from BL at Week 4 (n=96, 100, 92, 91) | -1.4 (0.7) | -1.1 (0.8) | 0.3 (0.8) | -1.8 (0.8)
  Change from BL at Week 6 (n=91, 98, 88, 84) | -1.5 (0.8) | -0.9 (0.8) | -0.8 (0.9) | -1.9 (0.9)
  Change from BL at Week 8 (n=94, 91, 91, 80) | -1.4 (0.9) | -0.9 (0.8) | -0.7 (0.8) | -2.4 (0.8)
  Change from BL at Week 10 (n=51, 66, 51, 50) | -0.8 (1.2) | -1.1 (1.1) | -1.3 (0.9) | -3.4 (1.1)
  Change from BL at Week 12 (n=82, 83, 87, 79) | -1.3 (0.9) | -2.0 (0.9) | -0.7 (0.8) | -1.8 (1.0)
  Change from BL at Week 14 (n=65, 72, 66, 62) | -2.5 (0.9) | -2.4 (1.1) | -2.4 (1.0) | -2.7 (1.0)
  Change from BL at Week 16 (n=87, 87, 81, 72) | -1.5 (0.9) | -0.5 (0.8) | -0.1 (0.9) | -2.1 (1.0)
  Change from BL at Week 18 (n=73, 69, 76, 66) | -2.3 (1.0) | -1.6 (0.9) | -1.9 (0.9) | -2.1 (1.1)
  Change from BL at Week 20 (n=84, 80, 76, 73) | -2.2 (0.9) | -1.8 (0.9) | -1.9 (1.0) | -2.2 (1.0)
  Change from BL at Week 22 (n=78, 73, 76, 64) | -3.0 (0.9) | -2.0 (0.9) | -2.5 (0.9) | -1.7 (1.1)
  Change from BL at Week 24 (n=84, 83, 77, 75) | -1.5 (1.0) | -1.7 (0.8) | -2.3 (0.9) | -3.4 (1.0)
  Change from BL at Week 30 (n=79, 78, 79, 66) | -1.4 (0.9) | -2.2 (0.9) | -0.3 (0.9) | -2.8 (1.0)
  Change from BL at Week 37 (n=77, 74, 71, 66) | -0.4 (1.1) | -1.7 (0.9) | -0.6 (1.0) | -2.0 (1.0)
  Change from BL at Week 50 (n=70, 73, 73, 62) | -1.7 (1.2) | 0.3 (0.8) | -0.3 (1.0) | -0.6 (1.1)
  Change from BL at Week 63 (n=61, 66, 69, 56) | -0.1 (1.2) | -0.4 (1.0) | -0.0 (1.0) | -0.5 (1.2)
  Change from BL at Week 76 (n=53, 59, 64, 50) | -1.6 (1.2) | -2.0 (0.8) | 0.1 (1.1) | -0.3 (1.4)
  Change from BL at Week 89 (n=49, 58, 56, 44) | 0.4 (1.2) | -2.1 (1.0) | -1.6 (1.2) | -0.1 (1.4)
  Change from BL at Week 102 (n=42, 51, 51, 42) | -1.1 (1.3) | -2.0 (1.2) | -0.4 (1.2) | -1.2 (1.2)
  Change from BL at Week 115 (n=34, 43, 43, 37) | -0.9 (1.5) | -2.7 (1.3) | -1.1 (1.1) | -1.0 (1.5)
  Change from BL at Week 128 (n=31, 40, 41, 31) | -1.8 (1.5) | -3.7 (1.2) | 1.1 (1.3) | 1.0 (1.6)
  Change from BL at Week 141 (n=29, 40, 35, 29) | 0.9 (1.5) | -2.0 (1.5) | 1.1 (1.7) | 1.3 (1.8)
  Change from BL at Week 154 (n=27, 36, 33, 27) | 1.2 (1.7) | -0.8 (1.3) | 2.5 (1.5) | 1.3 (1.8)
  Change from BL at Week 167 (n=24, 33, 30, 27) | 0.8 (1.6) | 0.3 (1.4) | 2.4 (1.8) | -1.1 (1.8)
  Change from BL at Week 180 (n=21, 28, 28, 27) | 1.4 (1.6) | -2.0 (2.0) | 0.5 (1.7) | -0.8 (1.9)
  Change from BL at Week 193 (n=19, 26, 27, 24) | 0.8 (2.3) | -1.6 (2.0) | 0.5 (1.7) | -0.2 (2.3)
  Change from BL at Week 206 (n=17, 24, 24, 23) | 0.3 (3.1) | -0.6 (2.4) | 1.9 (1.6) | -0.2 (2.4)

27. Other Pre Specified Outcome: Changes From Baseline in Heart Rate During the ST + LT Period
Time Frame: as for outcome 25
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
beats per minute
  Change from BL at Week 2 (n=96, 100, 94, 89) | -0.1 (0.9) | -0.5 (0.8) | 0.2 (0.8) | 0.3 (0.9)
  Change from BL at Week 4 (n=96, 100, 92, 91) | 0.2 (0.9) | -1.1 (0.8) | 0.7 (0.7) | -0.1 (0.9)
  Change from BL at Week 6 (n=91, 98, 88, 84) | -1.5 (0.9) | -0.6 (0.8) | -0.6 (0.8) | 1.4 (1.0)
  Change from BL at Week 8 (n=94, 91, 91, 80) | -0.5 (0.9) | -0.9 (0.8) | 0.2 (0.8) | -0.2 (0.9)
  Change from BL at Week 10 (n=51, 66, 51, 49) | -0.2 (1.2) | -1.5 (0.9) | -1.0 (1.2) | 0.1 (1.3)
  Change from BL at Week 12 (n=82, 83, 87, 79) | 0.3 (1.0) | -1.2 (0.8) | 0.5 (0.9) | 0.8 (1.1)
  Change from BL at Week 14 (n=65, 72, 65, 62) | 0.1 (1.1) | -0.5 (0.9) | 0.6 (1.1) | 1.9 (1.1)
  Change from BL at Week 16 (n=87, 87, 81, 72) | -0.8 (0.9) | -1.5 (0.9) | -0.1 (0.9) | -0.1 (1.0)
  Change from BL at Week 18 (n=73, 69, 76, 66) | -0.0 (1.1) | -0.8 (1.1) | 1.5 (1.0) | 2.6 (1.0)
  Change from BL at Week 20 (n=84, 80, 76, 73) | 1.3 (0.9) | -1.5 (0.9) | 1.3 (0.9) | 0.8 (1.1)
  Change from BL at Week 22 (n=78, 73, 76, 64) | 0.1 (1.0) | -0.3 (0.9) | 0.9 (0.9) | 1.5 (1.0)
  Change from BL at Week 24 (n=84, 83, 77, 75) | -0.3 (1.1) | 0.1 (1.1) | -0.7 (0.9) | -0.4 (1.1)
  Change from BL at Week 30 (n=79, 78, 79, 66) | -0.1 (1.0) | -1.2 (1.1) | -0.7 (0.8) | -1.2 (1.3)
  Change from BL at Week 37 (n=77, 74, 71, 66) | -0.4 (1.0) | -1.4 (0.9) | 0.5 (1.0) | -0.9 (1.2)
  Change from BL at Week 50 (n=70, 73, 73, 62) | -0.1 (0.9) | -0.7 (1.1) | -0.2 (1.0) | -0.2 (1.2)
  Change from BL at Week 63 (n=62, 66, 69, 56) | -0.4 (1.1) | -2.5 (1.0) | 0.9 (1.1) | 0.6 (1.4)
  Change from BL at Week 76 (n=53, 59, 64, 50) | -0.3 (1.4) | -3.3 (1.1) | 0.4 (1.1) | 0.2 (1.6)
  Change from BL at Week 89 (n=49, 58, 56, 44) | -0.5 (1.4) | -1.5 (1.2) | -0.9 (1.1) | -0.3 (1.3)
  Change from BL at Week 102 (n=42, 51, 51, 42) | -2.8 (1.4) | -1.5 (1.4) | -0.1 (1.4) | -0.0 (1.6)
  Change from BL at Week 115 (n=34, 43, 43, 37) | -3.2 (1.7) | -2.3 (1.3) | 1.0 (1.6) | 0.8 (1.9)
  Change from BL at Week 128 (n=31, 40, 41, 31) | -2.1 (1.8) | -4.5 (1.6) | -0.7 (1.4) | 1.7 (1.8)
  Change from BL at Week 141 (n=29, 40, 35, 29) | -2.8 (1.4) | -3.5 (1.5) | -0.6 (1.6) | 0.9 (1.7)
  Change from BL at Week 154 (n=27, 36, 33, 27) | -2.0 (2.1) | -2.6 (1.6) | -1.3 (1.8) | -0.6 (2.0)
  Change from BL at Week 167 (n=24, 33, 30, 27) | -5.1 (1.9) | -0.8 (1.4) | -2.1 (2.4) | 0.5 (1.6)
  Change from BL at Week 180 (n=21, 28, 28, 27) | -3.1 (2.1) | -5.3 (1.8) | -2.0 (2.0) | -1.2 (1.4)
  Change from BL at Week 193 (n=19, 26, 27, 24) | -4.6 (2.4) | -4.2 (1.8) | -2.4 (2.0) | 1.1 (2.1)
  Change from BL at Week 206 (n=17, 24, 24, 23) | -5.3 (2.6) | -2.6 (1.9) | 0.0 (2.7) | -0.8 (2.1)

28. Other Pre Specified Outcome: Electrocardiogram (ECG) Tracings - Shift Table From Baseline (BL) to Selected Visits During ST + LT Treatment Period
Description: The normality/abnormality of the ECG tracing was determined by the investigator.
Time Frame: Baseline, Weeks 12, 24, 76, 102, 154, 206
Population: Treated participants; BL n=number of participants at baseline
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
participants
  Normal BL, Normal Week 12 (BL n=65, 66, 67, 47) | 57 | 56 | 59 | 43
  Normal BL, Abnormal Week 12 (BL n=65, 66, 67, 47) | 8 | 10 | 8 | 4
  Abnormal BL, Normal Week 12 (BL n=27, 32, 26, 43) | 6 | 6 | 9 | 15
  Abnormal BL, Abnormal Week 12(BL n=27, 32, 26, 43) | 21 | 26 | 17 | 28
  Normal BL, Normal Week 24 (BL n=53, 52, 47, 33) | 43 | 44 | 43 | 31
  Normal BL, Abnormal Week 24 (BL n=53, 52, 47, 33) | 10 | 8 | 4 | 2
  Abnormal BL, Normal Week 24 (BL n=19, 24, 21, 25) | 5 | 8 | 9 | 8
  Abnormal BL, Abnormal Week 24(BL n=19, 24, 21, 25) | 14 | 16 | 12 | 17
  Normal BL, Normal Week 76 (BL n=48, 49, 48, 36) | 37 | 44 | 40 | 30
  Normal BL, Abnormal Week 76 (BL n=48, 49, 48, 36) | 11 | 5 | 8 | 6
  Abnormal BL, Normal Week 76 (BL n=19, 23, 21, 27) | 8 | 8 | 6 | 13
  Abnormal BL, Abnormal Week 76(BL n=19, 23, 21, 27) | 11 | 15 | 15 | 14
  Normal BL, Normal Week 102 (BL n=32, 32, 36, 22) | 25 | 26 | 31 | 18
  Normal BL, Abnormal Week 102 (BL n=32, 32, 36, 22) | 7 | 6 | 5 | 4
  Abnormal BL, Normal Week 102 (BL n=12, 18, 17, 20) | 4 | 5 | 12 | 11
  Abnormal BL,Abnormal Week 102(BL n=12, 18, 17, 20) | 8 | 13 | 5 | 9
  Normal BL, Normal Week 154 (BL n=20, 21, 26, 15) | 16 | 17 | 23 | 14
  Normal BL, Abnormal Week 154 (BL n=20, 21, 26, 15) | 4 | 4 | 3 | 1
  Abnormal BL, Normal Week 154 (BL n=7, 16, 11, 13) | 4 | 4 | 5 | 7
  Abnormal BL, Abnormal Week 154(BL n=7, 16, 11, 13) | 3 | 12 | 6 | 6
  Normal BL, Normal Week 206 (BL n=15, 13, 20, 14) | 15 | 12 | 18 | 11
  Normal BL, Abnormal Week 206 (BL n=15, 13, 20, 14) | 0 | 1 | 2 | 3
  Abnormal BL, Normal Week 206 (BL n=4, 13, 8, 11) | 2 | 3 | 4 | 4
  Abnormal BL, Abnormal Week 206 (BL n=4, 13, 8, 11) | 2 | 10 | 4 | 7

29. Other Pre Specified Outcome: Overall Summary of Adverse Events During ST+LT Treatment Period - Open-Label Cohort
Description: as for outcome 13
Time Frame: AEs: up to last treatment day + 1 day or last visit; SAEs: up to last treatment day + 30 days or last visit + 30 days. Mean duration of exposure was 34 weeks.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
participants
  At Least 1 AE | 49
  At Least 1 Related AE | 9
  Deaths | 0
  At Least 1 SAE | 6
  At Least 1 Related SAE | 0
  Discontinuations Due to SAEs | 2
  Discontinuations Due to AEs | 5

30. Other Pre Specified Outcome: Marked Laboratory Abnormalities During ST + LT Treatment Period - Open-Label Cohort
Description: as for outcome 14
Time Frame: Lab assessments taken during and up to 14 days after the last dose of study drug during the ST + LT Treatment Period. Mean duration of exposure was 34 weeks.
Population: as for outcome 14
Measure: Number; unit: participants
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 102
participants
  Hemoglobin < 8 g/dL (n=64) | 0
  Hematocrit < 0.75 x pre-Rx (n=64) | 0
  Platelets < 50 x 10^9 c/L (n=64) | 0
  Platelets > 1.5 x ULN (n=64) | 0
  Leukocytes < 2 x 1000 c/µL (n=64) | 0
  Neutrophils+Bands <1x1000 c/uL (n=64) | 1
  Eosinophils >0.9x1000 c/µL (n=64) | 2
  Lymphocytes <=0.75x1000 c/uL (n=64) | 0
  ALP >3 x pre-Rx and >ULN (n=64) | 0
  ALP >1.5 x ULN (n=64) | 0
  AST >3 x ULN (n=64) | 1
  AST >5 x ULN (n=64) | 0
  AST >10 x ULN (n=64) | 0
  AST >20 x ULN (n=64) | 0
  ALT >3 x ULN (n=64) | 1
  ALT >5 x ULN (n=64) | 0
  ALT >10 x ULN (n=64) | 0
  ALT >20 x ULN (n=64) | 0
  Bilirubin Total >2mg/dL (n=64) | 1
  Bilirubin Total >1.5xULN (n=64) | 1
  Bilirubin Total >2xULN (n=64) | 0
  BUN >2 x pre-Rx and >ULN (n=64) | 2
  Creatinine >2.5 mg/dL (n=64) | 0
  Glucose, Serum Fasting < 50 mg/dL (n=1) | 0
  Glucose, Serum Fasting > 500 mg/dL (n=1) | 0
  Glucose, Serum Unspec. < 50 mg/dL (n=1) | 0
  Glucose, Serum Unspec. > 500 mg/dL (n=1) | 0
  Glucose, Plasma Fasting <50 mg/dL (n=64) | 0
  Glucose,Plasma Fasting >500 mg/dL (n=64) | 0
  Glucose, Plasma Unspec. <50 mg/dL (n=65) | 2
  Glucose,Plasma Unspec. >500 mg/dL (n=65) | 1
  Sodium,Serum Low (see above) (n=65) | 0
  Sodium,Serum High (see above) (n=65) | 2
  Potassium,Serum Low (see above) (n=65) | 0
  Potassium, Serum High (see above) (n=65) | 2
  Chloride < 90 mEq/L (n=65) | 1
  Chloride > 120 mEq/L (n=65) | 0
  Albumin < 0.9 LLN (n=64) | 0
  Creatine Kinase > 5 x ULN (n=64) | 0
  Uric Acid > 1.5 x ULN (n=0) | 0
  Protein Urine, >=2-4 (n=64) | 2
  Blood Urine, >=2-4 (n=64) | 4
  Red Blood Cells Urine >=2-4 (n=58) | 7
  White Blood Cells Urine >=2-4 (n=58) | 6

31. Other Pre Specified Outcome: All Reported Hypoglycemic Adverse Events During ST + LT Treatment Period
Description: Hypoglycemic Events are based upon the Saxagliptin Predefined List of Events, which included hypoglycemia, blood glucose decreased, and hypoglycemic unconsciousness.
Time Frame: as for outcome 13
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
participants | 9 | 11 | 10 | 9

32. Other Pre Specified Outcome: Confirmed Hypoglycemia During ST + LT Treatment Period
Description: 'Confirmed' = recorded on the hypoglycemia AE case report form page with a fingerstick glucose <= 50 mg/dL and associated symptoms
Time Frame: as for outcome 13
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Saxagliptin 2.5 mg | Saxagliptin 5 mg | Saxagliptin 10 mg | Placebo
Number analyzed (Participants) | 102 | 106 | 98 | 95
participants | 1 | 1 | 0 | 0

33. Other Pre Specified Outcome: All Reported Hypoglycemic Adverse Events During ST + LT Treatment Period - Open-Label Cohort
Description: as for outcome 31
Time Frame: as for outcome 29
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 102
participants | 2

34. Other Pre Specified Outcome: Confirmed Hypoglycemia During ST + LT Treatment Period - Open-Label Cohort
Description: as for outcome 32
Time Frame: as for outcome 29
Population: Treated participants
Measure: Number; unit: participants
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
participants | 0

35. Other Pre Specified Outcome: Electrocardiogram (ECG) Tracings - Shift Table From Baseline (BL) to Selected Visits During ST + LT Treatment Period - Open Label Cohort
Description: The normality/abnormality of the ECG tracing was determined by the investigator.
Time Frame: Baseline, Weeks 12, 24, 76, 102, 154, 206
Population: Treated participants; BL n=number of participants at baseline
Measure: Number; unit: participants
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
participants
  Normal BL, Normal Week 12 (BL n=23) | 19
  Normal BL, Abnormal Week 12 (BL n=23) | 4
  Abnormal BL, Normal Week 12 (BL n=18) | 5
  Abnormal BL, Abnormal Week 12 (BL n=18) | 13
  Normal BL, Normal Week 24 (BL n=10) | 8
  Normal BL, Abnormal Week 24 (BL n=10) | 2
  Abnormal BL, Normal Week 24 (BL n=6) | 2
  Abnormal BL, Abnormal Week 24(BL n=6) | 4
  Normal BL, Normal Week 76 (BL n=17) | 13
  Normal BL, Abnormal Week 76 (BL n=17) | 4
  Abnormal BL, Normal Week 76 (BL n=13) | 4
  Abnormal BL, Abnormal Week 76 (BL n=13) | 9
  Normal BL, Normal Week 102 (BL n=8) | 6
  Normal BL, Abnormal Week 102 (BL n=8) | 2
  Abnormal BL, Normal Week 102 (BL n=4) | 1
  Abnormal BL, Abnormal Week 102 (BL n=4) | 3
  Normal BL, Normal Week 154 (BL n=4) | 3
  Normal BL, Abnormal Week 154 (BL n=4) | 1
  Abnormal BL, Normal Week 154 (BL n=2) | 0
  Abnormal BL, Abnormal Week 154 (BL n=2) | 2
  Normal BL, Normal Week 206 (BL n=3) | 2
  Normal BL, Abnormal Week 206 (BL n=3) | 1
  Abnormal BL, Normal Week 206 (BL n=1) | 0
  Abnormal BL, Abnormal Week 206 (BL n=1) | 1

36. Other Pre Specified Outcome: Changes From Baseline in Systolic Blood Pressure During the ST + LT Period - Open Label Cohort
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
mmHg
  Change from BL at Week 2 (n=62) | -4.4 (1.3)
  Change from BL at Week 4 (n=59) | -3.8 (1.4)
  Change from BL at Week 6 (n=60) | -2.7 (1.5)
  Change from BL at Week 8 (n=49) | -5.1 (1.6)
  Change from BL at Week 10 (n=24) | -4.2 (2.8)
  Change from BL at Week 12 (n=47) | -4.9 (1.8)
  Change from BL at Week 14 (n=35) | -5.1 (2.0)
  Change from BL at Week 16 (n=46) | -1.9 (2.2)
  Change from BL at Week 18 (n=42) | -5.8 (2.0)
  Change from BL at Week 20 (n=45) | -3.6 (2.0)
  Change from BL at Week 22 (n=44) | -4.0 (2.1)
  Change from BL at Week 24 (n=44) | -4.3 (2.1)
  Change from BL at Week 30 (n=40) | -4.8 (1.8)
  Change from BL at Week 37 (n=35) | -4.7 (1.8)
  Change from BL at Week 50 (n=36) | -1.6 (2.1)
  Change from BL at Week 63 (n=26) | -0.7 (2.7)
  Change from BL at Week 76 (n=24) | -1.9 (2.1)
  Change from BL at Week 89 (n=23) | -4.0 (2.6)
  Change from BL at Week 102 (n=15) | 0.9 (2.4)
  Change from BL at Week 115 (n=13) | -6.6 (3.6)
  Change from BL at Week 128 (n=11) | -5.6 (4.3)
  Change from BL at Week 141 (n=10) | -7.2 (4.4)
  Change from BL at Week 154 (n=10) | 5.7 (4.7)
  Change from BL at Week 167 (n=10) | -2.2 (4.4)

37. Other Pre Specified Outcome: Changes From Baseline in Diastolic Blood Pressure During the ST + LT Period - Open Label Cohort
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
mmHg
  Change from BL at Week 2 (n=62) | -3.7 (0.9)
  Change from BL at Week 4 (n=59) | -1.7 (1.0)
  Change from BL at Week 6 (n=60) | -2.8 (1.0)
  Change from BL at Week 8 (n=49) | -2.0 (1.1)
  Change from BL at Week 10 (n=24) | -1.0 (2.0)
  Change from BL at Week 12 (n=47) | -3.7 (1.4)
  Change from BL at Week 14 (n=35) | -4.5 (1.7)
  Change from BL at Week 16 (n=46) | -2.8 (1.2)
  Change from BL at Week 18 (n=42) | -3.3 (1.1)
  Change from BL at Week 20 (n=45) | -2.1 (1.2)
  Change from BL at Week 22 (n=44) | -2.8 (1.5)
  Change from BL at Week 24 (n=44) | -3.4 (1.3)
  Change from BL at Week 30 (n=40) | -3.8 (1.5)
  Change from BL at Week 37 (n=35) | -2.0 (1.4)
  Change from BL at Week 50 (n=36) | -1.3 (1.4)
  Change from BL at Week 63 (n=26) | -0.9 (1.8)
  Change from BL at Week 76 (n=24) | -1.0 (2.0)
  Change from BL at Week 89 (n=23) | -2.6 (1.9)
  Change from BL at Week 102 (n=15) | 1.0 (3.0)
  Change from BL at Week 115 (n=13) | -4.1 (2.5)
  Change from BL at Week 128 (n=11) | -3.7 (2.8)
  Change from BL at Week 141 (n=10) | -6.0 (2.6)
  Change from BL at Week 154 (n=10) | -0.5 (2.7)
  Change from BL at Week 167 (n=10) | -2.5 (2.9)

38. Other Pre Specified Outcome: Changes From Baseline in Heart Rate During the ST + LT Period - Open Label Cohort
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 30, 37, 50, 63, 76, 89, 102, 115, 128, 141, 154, 167
Population: Treated participants; n=number of treated participants with measurement at time point
Measure: Mean (Standard Error); unit: beats per minute
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees)
Number analyzed (Participants) | 66
beats per minute
  Change from BL at Week 2 (n=62) | -0.8 (1.0)
  Change from BL at Week 4 (n=59) | -0.4 (1.1)
  Change from BL at Week 6 (n=60) | -0.3 (1.0)
  Change from BL at Week 8 (n=49) | -0.7 (1.5)
  Change from BL at Week 10 (n=23) | -1.8 (2.1)
  Change from BL at Week 12 (n=47) | -3.0 (1.1)
  Change from BL at Week 14 (n=34) | -2.0 (1.4)
  Change from BL at Week 16 (n=46) | -0.7 (1.1)
  Change from BL at Week 18 (n=42) | -2.0 (1.3)
  Change from BL at Week 20 (n=45) | 1.6 (1.1)
  Change from BL at Week 22 (n=43) | -0.4 (1.2)
  Change from BL at Week 24 (n=44) | -0.4 (1.5)
  Change from BL at Week 30 (n=40) | 0.6 (1.3)
  Change from BL at Week 37 (n=35) | -1.6 (1.6)
  Change from BL at Week 50 (n=36) | -2.9 (1.3)
  Change from BL at Week 63 (n=26) | -3.0 (1.6)
  Change from BL at Week 76 (n=24) | -0.4 (2.5)
  Change from BL at Week 89 (n=23) | -1.3 (1.8)
  Change from BL at Week 102 (n=15) | -0.3 (1.6)
  Change from BL at Week 115 (n=13) | 1.7 (1.6)
  Change from BL at Week 128 (n=11) | -1.6 (3.6)
  Change from BL at Week 141 (n=10) | -3.4 (1.7)
  Change from BL at Week 154 (n=10) | -1.5 (2.6)
  Change from BL at Week 167 (n=10) | -1.9 (3.3)

ADVERSE EVENTS:
Arm/Group | Open-Label Treatment Cohort (Direct Enrollees) | Placebo | Saxagliptin 10 mg | Saxagliptin 2.5 mg | Saxagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 6/66 | 11/95 | 9/98 | 11/102 | 18/106
Other Adverse Events (participants affected / at risk) | 39/66 | 63/95 | 69/98 | 72/102 | 77/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Treatment Cohort (Direct Enrollees) (N=66) | Placebo (N=95) | Saxagliptin 10 mg (N=98) | Saxagliptin 2.5 mg (N=102) | Saxagliptin 5 mg (N=106)
TACHYCARDIA (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
ANGINA UNSTABLE (Cardiac disorders) | 0 | 1 | 0 | 1 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
AORTIC VALVE STENOSIS (Cardiac disorders) | 0 | 0 | 1 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 0 | 0 | 2 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
HYPOTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 0 | 1
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 | 1 | 0 | 0 | 0
ADRENAL MASS (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1
GALLBLADDER POLYP (Hepatobiliary disorders) | 0 | 1 | 0 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 1 | 0 | 2 | 1
SCIATICA (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
VASCULAR HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
IVTH NERVE PARALYSIS (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
INTESTINAL MASS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
ABDOMINAL TENDERNESS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
GANGRENE (Infections and infestations) | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 1 | 1 | 0 | 2 | 0
CELLULITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 2
HEPATITIS C (Infections and infestations) | 0 | 0 | 0 | 1 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
TUBERCULOSIS (Infections and infestations) | 0 | 0 | 1 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
HAEMATOMA INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 1
NEPHROLITHIASIS (Renal and urinary disorders) | 1 | 1 | 0 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
RASH (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
TESTICULAR PAIN (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0
WOUND (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 1 | 1 | 1 | 0
NON-CARDIAC CHEST PAIN (General disorders) | 0 | 0 | 0 | 0 | 1
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1
BRAIN NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1 | 0
CERVIX CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1 | 0
RENAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-Label Treatment Cohort (Direct Enrollees) (N=66) | Placebo (N=95) | Saxagliptin 10 mg (N=98) | Saxagliptin 2.5 mg (N=102) | Saxagliptin 5 mg (N=106)
HYPERTENSION (Vascular disorders) | 2 | 8 | 3 | 5 | 7
INSOMNIA (Psychiatric disorders) | 1 | 3 | 3 | 3 | 6
DEPRESSION (Psychiatric disorders) | 3 | 3 | 6 | 2 | 7
HEADACHE (Nervous system disorders) | 8 | 16 | 16 | 7 | 13
DIZZINESS (Nervous system disorders) | 5 | 8 | 3 | 4 | 9
NAUSEA (Gastrointestinal disorders) | 6 | 6 | 4 | 7 | 6
VOMITING (Gastrointestinal disorders) | 3 | 3 | 1 | 4 | 7
DIARRHOEA (Gastrointestinal disorders) | 4 | 8 | 10 | 14 | 8
TOOTHACHE (Gastrointestinal disorders) | 0 | 5 | 2 | 3 | 3
CONSTIPATION (Gastrointestinal disorders) | 1 | 5 | 3 | 3 | 5
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2 | 1 | 2 | 7
INFLUENZA (Infections and infestations) | 4 | 6 | 15 | 11 | 9
SINUSITIS (Infections and infestations) | 2 | 5 | 10 | 9 | 8
BRONCHITIS (Infections and infestations) | 1 | 6 | 5 | 2 | 5
PHARYNGITIS (Infections and infestations) | 2 | 6 | 6 | 4 | 6
NASOPHARYNGITIS (Infections and infestations) | 8 | 12 | 14 | 11 | 13
URINARY TRACT INFECTION (Infections and infestations) | 6 | 8 | 10 | 8 | 14
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 15 | 14 | 12 | 16
RASH (Skin and subcutaneous tissue disorders) | 4 | 2 | 5 | 7 | 8
CONTUSION (Injury, poisoning and procedural complications) | 1 | 2 | 2 | 7 | 2
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 11 | 5 | 4 | 12
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 4 | 7 | 16 | 8 | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 6 | 9 | 9 | 8
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 5 | 9 | 6 | 4 | 5
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 6 | 5 | 4
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 3 | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.